CLINICAL TRIAL: NCT00261443
Title: Efficacy of Aripiprazole in Combination With Lithium or Valproate in the Long-Term Maintenance Treatment of Bipolar I Disorder in Outpatients Partially Nonresponsive to Lithium or Valproate Monotherapy
Brief Title: A Study of Aripiprazole (Abilify) in Patients With Bipolar Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-189
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Results first posted 2011-04-27 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder with a recent manic or mixed episode
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Valproic Acid; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Placebo Comparator): /Active Comparator
  Interventions: Drug: Lithium or Valproate with placebo (PBO)
- A2 (Experimental)
  Interventions: Drug: Lithium or Valproate with Aripiprazole

INTERVENTIONS:
Drug: Lithium or Valproate with placebo (PBO) — Tablets, Oral, once daily
  lithium 250-2100 mg/day
  valproate 250-2500mg/day
  Placebo once daily
  Arms: A1
Drug: Lithium or Valproate with Aripiprazole — Tablets, Oral, once daily, 52 weeks post randomization (Pre-Randomization Phases 13-24 weeks)
  lithium 250-2100 mg/day
  valproate 250-2500mg/day
  aripiprazole 15-30 mg/day
  Other Names: Abilify; BMS-337039
  Arms: A2

SUMMARY:
The purpose of this clinical research study is to learn if outpatients with bipolar mania who are partially nonresponsive to lithium or valproate monotherapy can achieve stable symptoms on a combination treatment of aripiprazole plus lithium or valproate.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > or = to 18 years of age meeting Diagnostic and Statistical Manual for Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for bipolar I disorder, currently experiencing a manic or mixed episode with a history of one or more manic or mixed episodes or sufficient severity to require hospitalization and/or treatment with a mood stabilizer or antipsychotic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1270 (Actual)
Dates: Start 2005-09; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (76):
- United States (29):
  - Tuscaloosa Va Medical Center, Tuscaloosa, Alabama
  - Pravin Kansagra, M.D., Anaheim, California
  - Psychopharmacology Research Network Of Torrance, Cerritos, California
  - Atp Clinical Research, Inc., Costa Mesa, California
  - Us Clinical Research Centers, Llc, Costa Mesa, California
  - Va Long Beach Healthcare System, Long Beach, California
  - Synergy Clinical Research Center, National City, California
  - University Of California, Irvine Medical Center, Orange, California
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - University Of South Florida, Tampa, Florida
  - Carman Research, Smyrna, Georgia
  - University Of Massachusetts Medical School, Worcester, Massachusetts
  - Psych Care Consultants Research, St Louis, Missouri
  - Cns Research Institute, P.C., Clementon, New Jersey
  - Neuropsychiatric Research Associates, New York, New York
  - Behavioral Medical Research Of Staten Island, Staten Island, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Psychiatry And Clinical Research, Raleigh, North Carolina
  - Rakesh Ranjan, Md & Associates, Inc., Beachwood, Ohio
  - University Of Cincinnati Medical Center, Cincinnati, Ohio
  - Metro Health Medical Center, Cleveland, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Portland Va Medical Center, Portland, Oregon
  - Senior Adults Specialty Research, Inc., Austin, Texas
  - Futuresearch Trials, Dallas, Texas
  - Insite Clinical Research, DeSoto, Texas
  - Red Oak Psychiatry Associates, Pa, Houston, Texas
  - University Of Utah School Of Medicine, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
- Brazil (5):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Aparecida de Goinia, Goiás
  - Local Institution, Pelotas, Rio Grande do Sul
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Bulgaria (2):
  - Local Institution, Burgas
  - Local Institution, Rousse
- Croatia (4):
  - Local Institution, Rijeka
  - Local Institution, Split
  - Local Institution, Zadar
  - Local Institution, Zagreb
- Czechia (5):
  - Local Institution, Brno
  - Local Institution, Havířov
  - Local Institution, Litoměřice
  - Local Institution, Prague
  - Local Institution, Přerov
- France (9):
  - Local Institution, Nantes, Cedex 01
  - Local Institution, Dole
  - Local Institution, Hénin-Beaumont
  - Local Institution, Jonzac
  - Local Institution, La Seyne-sur-Mer
  - Local Institution, Marseille
  - Local Institution, Nantes
  - Local Institution, Nîmes
  - Local Institution, Rennes
- India (11):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Kalyan (West), Maharashtra
  - Local Institution, Nāgūr, Maharashtra
  - Local Institution, Pune, Maharashtra
  - Local Institution, Mangalore, Manipal
  - Local Institution, Mumbai, Sion (W)
  - Local Institution, Delhi
  - Local Institution, Hyderabad
  - Local Institution, Mumbai
  - Local Institution, New Delhi
- Russia (6):
  - Local Institution, Izhevsk
  - Local Institution, Moscow
  - Local Institution, Nizhny Novgorod
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Tomsk
- South Africa (5):
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Berea, KwaZulu-Natal
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Paarl, Western Cape

REFERENCES:
- [Derived] Marcus R, Khan A, Rollin L, Morris B, Timko K, Carson W, Sanchez R. Efficacy of aripiprazole adjunctive to lithium or valproate in the long-term treatment of patients with bipolar I disorder with an inadequate response to lithium or valproate monotherapy: a multicenter, double-blind, randomized study. Bipolar Disord. 2011 Mar;13(2):133-44. doi: 10.1111/j.1399-5618.2011.00898.x. PMID 21443567

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-Randomized Participants: Phase 1 (2 to 8 Week Screening, Washout and Confirmation of Partial Nonresponse Phase): lithium: 0.6-1.0 mmol/L or valproate 50-125 µg/ml. Phase 2 (13 to 24 Week Stability and Maintenance of Stability Phase): 10-mg, 15-mg, or 30-mg doses of aripiprazole and lithium: 0.6-1.0 mmol/L or valproate 50-125 µg/ml.
- Placebo: Phase 3 (52 Week Assessment of Relapse Phase): matching placebo oral tablets and lithium: 0.6-1.0 mmol/L or valproate 50-125 µg/ml.
- Aripiprazole: Phase 3 (52 Week Assessment of Relapse Phase): 10-mg, 15-mg, or 30-mg doses of aripiprazole and lithium: 0.6-1.0 mmol/L or valproate 50-125 µg/ml.
Period: 1: Confirmation of Partial Nonresponse
Arm/Group | Pre-Randomized Participants | Placebo | Aripiprazole
Started | 1270 | 0 | 0
Completed | 686 | 0 | 0
Not Completed | 584 | 0 | 0
Not completed — Adverse Event | 33 | 0 | 0
Not completed — Withdrawal by Subject | 93 | 0 | 0
Not completed — Lost to Follow-up | 111 | 0 | 0
Not completed — Poor/Noncompliance | 23 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Subject No Longer Met Study Criteria | 307 | 0 | 0
Not completed — Other Reasons | 16 | 0 | 0
Period: 2: Stability & Maintenance of Stability
Arm/Group | Pre-Randomized Participants | Placebo | Aripiprazole
Started | 686 | 0 | 0
Completed | 346 | 0 | 0
Not Completed | 340 | 0 | 0
Not completed — Lack of Efficacy | 43 | 0 | 0
Not completed — Adverse Event | 93 | 0 | 0
Not completed — Withdrawal by Subject | 65 | 0 | 0
Not completed — Lost to Follow-up | 59 | 0 | 0
Not completed — Poor/Noncompliance | 33 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — subject No Longer Met Study Criteria | 32 | 0 | 0
Not completed — Administrative Reason by Sponsor | 1 | 0 | 0
Not completed — Other Reasons | 13 | 0 | 0
Period: 3: Assessment of Relapse
Arm/Group | Pre-Randomized Participants | Placebo | Aripiprazole
Started | 0 | 169 | 168
Completed | 0 | 89 | 103
Not Completed | 0 | 80 | 65
Not completed — Lack of Efficacy | 0 | 31 | 14
Not completed — Adverse Event | 0 | 15 | 19
Not completed — Withdrawal by Subject | 0 | 14 | 15
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 7 | 6
Not completed — Poor/Noncompliance | 0 | 5 | 3
Not completed — Pregnancy | 0 | 2 | 1
Not completed — Subject No Longer Meets Study Criteria | 0 | 2 | 1
Not completed — Administrative Reason By Sponsor | 0 | 0 | 2
Not completed — Other Reasons | 0 | 4 | 3
Period: 4: Extension Phase
Arm/Group | Pre-Randomized Participants | Placebo | Aripiprazole
Started | 0 | 19 | 23
Completed | 0 | 16 | 21
Not Completed | 0 | 3 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Phase 3 (52 Week Assessment of Relapse Phase): matching placebo oral tablets and 250-mg and 300-mg oral lithium tablets or 250-mg Depakote/valproic acid oral tablets
- Aripiprazole: Phase 3 (52 Week Assessment of Relapse Phase): aripiprazole 10-mg and 15-mg oral tablets and 250-mg and 300-mg oral lithium tablets or 250-mg Depakote/valproic acid oral tablets
- Total: Total of all reporting groups
Arm/Group | Placebo | Aripiprazole | Total
Number analyzed (Participants) | 169 | 168 | 337
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (12.29) | 39.2 (12.43) | 39.0 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 87 | 185
  Male | 71 | 81 | 152
Race/Ethnicity, Customized [Number; unit: participants]
  White | 112 | 118 | 230
  Black/African American | 19 | 12 | 31
  Asian | 33 | 34 | 67
  Other | 5 | 4 | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic/Latino | 3 | 5 | 8
  Not Hispanic or Latino | 55 | 56 | 111
  Non-US | 111 | 107 | 218
Region of Enrollment [Number; unit: participants]
  France | 8 | 9 | 17
  United States | 58 | 61 | 119
  Czech Republic | 18 | 14 | 32
  Brazil | 28 | 27 | 55
  Croatia | 3 | 4 | 7
  Russian Federation | 17 | 15 | 32
  South Africa | 4 | 4 | 8
  India | 33 | 34 | 67
Body Mass Index (BMI) Category [Number; unit: Participants] — BMI is defined as weight in kilograms divided by the square of height in meters.
  Participants
    <18.5 kg/m^2 | 5 | 0 | 5
    18.5 kg/m^2 to <25 kg/m^2 | 58 | 49 | 107
    25 kg/m^2 to <30 kg/m^2 | 50 | 63 | 113
    >= 30 kg/m^2 | 56 | 56 | 112
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is defined as weight in kilograms divided by the square of height in meters.
  kg/m^2 | 28.7 (7.72) | 28.5 (6.00) | 28.6 (6.90)
CGI-BP Change from Preceding Phase Score (Depression) [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change in patients with bipolar disorder. Patients are rated on Change from Preceding Phase (mania, depression and overall bipolar illness) items (also a 7-point scale (1 to 7), with 1 being very much improved and 7 being very much worse).
  units on a scale | 3.0 (1.34) | 3.0 (1.31) | 3.0 (1.32)
CGI-BP Change from Preceding Phase Score (Mania) [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change in patients with bipolar disorder. Patients are rated on Change from Preceding Phase (mania, depression and overall bipolar illness) items (also a 7-point scale (1 to 7), with 1 being very much improved and 7 being very much worse).
  units on a scale | 1.6 (0.81) | 1.4 (0.63) | 1.5 (0.72)
CGI-BP Change from Preceding Phase Score (Overall) [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change in patients with bipolar disorder. Patients are rated on Change from Preceding Phase (mania, depression and overall bipolar illness) items (also a 7-point scale (1 to 7), with 1 being very much improved and 7 being very much worse).
  units on a scale | 1.6 (0.85) | 1.5 (0.69) | 1.6 (0.77)
CGI-BP Severity of Illness Score (Depression) [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change in patients with bipolar disorder. Patients are rated on Severity of Illness (mania, depression, and overall bipolar illness) items (a 7-point scale from 1 to 7, with 1 being normal, not ill and 7 being very severely ill).
  units on a scale | 1.3 (0.57) | 1.4 (0.70) | 1.4 (0.64)
CGI-BP Severity of Illness Score (Mania) [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change in patients with bipolar disorder. Patients are rated on Severity of Illness (mania, depression, and overall bipolar illness) items (a 7-point scale from 1 to 7, with 1 being normal, not ill and 7 being very severely ill).
  units on a scale | 1.5 (0.72) | 1.5 (0.72) | 1.5 (0.72)
CGI-BP Severity of Illness Score (Overall) [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change in patients with bipolar disorder. Patients are rated on Severity of Illness (mania, depression, and overall bipolar illness) items (a 7-point scale from 1 to 7, with 1 being normal, not ill and 7 being very severely ill).
  units on a scale | 1.6 (0.76) | 1.7 (0.83) | 1.6 (0.79)
Montgomery Åsberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — MADRS consists of 10-items, ordinal rating scale The possible total scores are from 0 to 60 (0=no symptoms; 60=most severe symptoms). Change from baseline=postbaseline score - baseline score. A negative change score indicates improvement.
  units on a scale | 3.7 (3.45) | 4.1 (3.82) | 3.9 (3.64)
Weight [Mean (Standard Deviation); unit: kg] | 81.3 (25.11) | 80.6 (18.89) | 81.0 (22.20)
Young-Mania Rating Scale (Y-MRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The Y-MRS consists of 11 items: 1) Elevated Mood, 2) Increased Motor Activity -Energy, 3) Sexual Interest, 4) Sleep, 5) Irritability, 6) Speech (Rate and Amount), 7) Language -Thought Disorder, 8) Content, 9) Disruptive-Aggressive Behavior, 10) Appearance, 11) Insight. Seven items are rated on a 0 to 4 scale, while 4 items (items 5, 6, 8 and 9) are rated on a 0 to 8 scale (twice the weight of the other items.) For all items, 0 is the "best" rating and 4 or 8 is the "worst" rating. Total Score is the sum of the ratings for all 11 items. The possible Total Scores are from 0 to 60.
  units on a scale | 4.1 (3.31) | 4.1 (3.56) | 4.1 (3.43)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Not Experiencing Relapse to Any Mood Episode Through Week 52, Phase 3
Description: Kaplan-Meier estimated survival rate. Criteria for relapse include one or more of the following: hospitalization for a manic, mixed or depressive episode; serious adverse event of worsening disease under study accompanied by a Y-MRS > 16 and/or a MADRS > 16; discontinuation due to lack of efficacy as determined by the investigator accompanied by a Y-MRS > 16 and/or a MADRS > 16.
Time Frame: Week 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 of Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: Randomized Sample; n=number of participants at risk at each time point
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 169 | 168
proportion of participants
  Proportion at Week 0 (n=169, 168) | 1.00 | 1.00
  Proportion at Week 4 (n=153, 148) | 0.95 | 0.96
  Proportion at Week 8 (n=148, 139) | 0.93 | 0.94
  Proportion at Week 12 (n=142, 133) | 0.90 | 0.93
  Proportion at Week 16 (n=131, 130) | 0.87 | 0.92
  Proportion at Week 20 (n=122, 128) | 0.83 | 0.91
  Proportion at Week 24 (n=113, 125) | 0.81 | 0.89
  Proportion at Week 28 (n=105, 121) | 0.77 | 0.89
  Proportion at Week 32 (n=102, 114) | 0.76 | 0.84
  Proportion at Week 36 (n=99, 111) | 0.75 | 0.84
  Proportion at Week 40 (n=95, 110) | 0.73 | 0.84
  Proportion at Week 44 (n=91,107) | 0.73 | 0.84
  Proportion at Week 48 (n=88, 98) | 0.71 | 0.83
  Proportion at Week 52 (n=5, 8) | 0.71 | 0.83
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Test type: Superiority or Other; p = 0.014, Stratified Log-rank Test — Stratified Log-rank Test, controlling for type of mood stabilizer and type of mood episode; Hazard Ratio (HR) = 0.544, 95% CI 2-sided [0.332 to 0.893] — Cox proportional hazards model, with type of mood stabilizer and type of index mood episode as stratification factors, and treatment group as covariate

2. Secondary Outcome: Baseline and Adjusted Mean Change From Baseline in Clinical Global Impression Scale for Bipolar Disorder (CGI-BP) Severity of Illness Score (Mania) Through Phase 3
Description: Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change from baseline in patients with bipolar disorder. Patients are rated on mania, depression and overall bipolar illness items on a 7-point scale [1 to 7], with 1 being normal and 7 being very severely ill). A negative change score signifies improvement.
Time Frame: Baseline (end of Phase 2), 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: LOCF data set, phase 3 efficacy sample; n=number of participants evaluated at given time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Mean Baseline (n=164, 162) | 1.54 (0.059) | 1.54 (0.058)
  Mean Change from Baseline to Week 4 (n=160, 162) | 0.01 (0.052) | 0.05 (0.050)
  Mean Change from Baseline to Week 8 (n=164, 162) | 0.05 (0.054) | 0.01 (0.053)
  Mean Change from Baseline to Week 12 (n=164, 162) | 0.12 (0.063) | 0.07 (0.062)
  Mean Change from Baseline to Week 16 (n=164, 162) | 0.19 (0.064) | 0.07 (0.063)
  Mean Change from Baseline to Week 20 (n=164, 162) | 0.23 (0.071) | 0.07 (0.070)
  Mean Change from Baseline to Week 24 (n=164, 162) | 0.25 (0.074) | 0.05 (0.073)
  Mean Change from Baseline to Week 28 (n=164, 162) | 0.31 (0.082) | 0.10 (0.080)
  Mean Change from Baseline to Week 32 (n=164, 162) | 0.27 (0.078) | 0.08 (0.076)
  Mean Change from Baseline to Week 36 (n=164, 162) | 0.30 (0.079) | 0.05 (0.078)
  Mean Change from Baseline to Week 40 (n=164, 162) | 0.27 (0.080) | 0.05 (0.079)
  Mean Change from Baseline to Week 44 (n=164, 162) | 0.33 (0.082) | 0.06 (0.080)
  Mean Change from Baseline to Week 48 (n=164, 162) | 0.33 (0.082) | 0.05 (0.081)
  Mean Change from Baseline to Week 52 (n=164, 162) | 0.32 (0.083) | 0.04 (0.082)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Baseline Comparison; Test type: Superiority or Other; p = 0.911, ANOVA/ANCOVA — ANOVA model, controlling for treatment, mood stabilizer, and index mood episode used for baseline. ANCOVA model, controlling for treatment, mood stabilizer, index mood episode, and baseline value used for mean change from baseline; Means, difference in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.01, 95% CI 2-sided [-0.16 to 0.15]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 4 Comparison; Test type: Superiority or Other; p = 0.557, ANOVA/ANCOVA — Mean change from baseline: ANOVA controlling for treatment, mood stabilizer, type of index mood episode, baseline value. Mean change from preceding phase: ANCOVA controlling for treatment, mood stabilizer, type of index mood episode, baseline CGI-BP; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = 0.04, 95% CI 2-sided [-0.09 to 0.18]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 8 Comparison; Test type: Superiority or Other; p = 0.596, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.04, 95% CI 2-sided [-0.18 to 0.10]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 12 Comparison; Test type: Superiority or Other; p = 0.522, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.05, 95% CI 2-sided [-0.22 to 0.11]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 16 Comparison; Test type: Superiority or Other; p = 0.142, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.13, 95% CI 2-sided [-0.30 to 0.04]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 20 Comparison; Test type: Superiority or Other; p = 0.092, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.16, 95% CI 2-sided [-0.35 to 0.03]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 24 Comparison; Test type: Superiority or Other; p = 0.039, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.20, 95% CI 2-sided [-0.40 to -0.01]
Statistical Analysis 8: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 28 Comparison; Test type: Superiority or Other; p = 0.050, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.21, 95% CI 2-sided [-0.43 to 0.00]
Statistical Analysis 9: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 32 Comparison; Test type: Superiority or Other; p = 0.064, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.19, 95% CI 2-sided [-0.40 to 0.01]
Statistical Analysis 10: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 36 Comparison; Test type: Superiority or Other; p = 0.017, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.25, 95% CI 2-sided [-0.46 to -0.05]
Statistical Analysis 11: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 40 Comparison; Test type: Superiority or Other; p = 0.039, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.22, 95% CI 2-sided [-0.43 to -0.01]
Statistical Analysis 12: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 44 Comparison; Test type: Superiority or Other; p = 0.015, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.27, 95% CI 2-sided [-0.48 to -0.05]
Statistical Analysis 13: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 48 Comparison; Test type: Superiority or Other; p = 0.009, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.29, 95% CI 2-sided [-0.50 to -0.07]
Statistical Analysis 14: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 52 Comparison; Test type: Superiority or Other; p = 0.013, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.28, 95% CI 2-sided [-0.50 to -0.06]

3. Secondary Outcome: Proportion of Participants Not Experiencing Relapse of Manic Episode Through Phase 3
Description: Kaplan-Meier estimated survival rate. Criteria for relapse include one or more of the following: relapse is defined as any of the following events accompanied by a Young-Mania Rating Scale (Y-MRS) >16 and/or a Montgomery Åsberg Depression Rating Scale (MADRS) >16; serious adverse event of worsening disease, or discontinuation by the investigator for lack of efficacy. A hospitalization for a manic, mixed, or depressive episode does meet the criteria for relapse, however does not require an accompanying Y-MRS and/or MADRS score >16.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 of phase 3
Population: Randomized sample, n=number of participants at risk at given time point
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 169 | 168
proportion of participants
  Proportion at Week 0 (n=169,168) | 1.00 | 1.00
  Proportion at Week 4 (n=153,148) | 0.99 | 0.99
  Proportion at Week 8 (n=148,139) | 0.99 | 0.98
  Proportion at Week 12 (n=142,133) | 0.97 | 0.97
  Proportion at Week 16 (n=132,130) | 0.95 | 0.97
  Proportion at Week 20 (n=122,128) | 0.93 | 0.97
  Proportion at Week 24 (n=113,125) | 0.91 | 0.97
  Proportion at Week 28 (n=105,121) | 0.90 | 0.97
  Proportion at Week 32 (n=102,115) | 0.89 | 0.95
  Proportion at Week 36 (n=99, 111) | 0.88 | 0.95
  Proportion at Week 40 (n=95,110) | 0.87 | 0.95
  Proportion at Week 44 (n=91,107) | 0.86 | 0.95
  Proportion at Week 48 (n=88, 98) | 0.85 | 0.95
  Proportion at Week 52 (n=5, 8) | 0.85 | 0.95
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Test type: Superiority or Other; p = 0.013, Stratified Log-rank Test — Stratified Log-rank Test, controlling for type of mood stabilizer and type of index mood episode; Hazard Ratio (HR) = 0.348, 95% CI 2-sided [0.146 to 0.829] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Proportion of Participants Not Experiencing Relapse of Depressive Episode Through Week 52 During Phase 3
Description: Kaplan Meier estimated survival rate. Relapse is defined as any of the following events accompanied by a YMRS > 16 and/or a MADRS > 16; serious adverse event of worsening disease, or discontinuation by the investigator for lack of efficacy. A hospitalization for a manic, mixed, or depressive episode does meet the criteria for relapse, however does not require an accompanying Y-MRS and/or MADRS score > 16.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 of phase 3
Population: Randomized sample, n=number of participants at risk at given time point
Measure: Number; unit: proportion of participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 169 | 168
proportion of participants
  Proportion at Week 0 (n=169, 168) | 1.00 | 1.00
  Proportion at Week 4 (n=153, 148) | 0.96 | 0.98
  Proportion at Week 8 (n=148, 139) | 0.94 | 0.97
  Proportion at Week 12 (n=142, 133) | 0.94 | 0.97
  Proportion at Week 16 (n=132, 130) | 0.93 | 0.96
  Proportion at Week 20 (n=123, 128) | 0.92 | 0.96
  Proportion at Week 24 (n=115, 125) | 0.92 | 0.95
  Proportion at Week 28 (n=107, 121) | 0.89 | 0.95
  Proportion at Week 32 (n=104, 114) | 0.89 | 0.91
  Proportion at Week 36 (n=101, 111) | 0.89 | 0.91
  Proportion at Week 40 (n=98, 110) | 0.88 | 0.91
  Proportion at Week 44 (n=94, 107) | 0.88 | 0.91
  Proportion at Week 48 (n=91, 98) | 0.87 | 0.90
  Proportion at Week 52 (n=6, 8) | 0.87 | 0.90
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Test type: Superiority or Other; p = 0.384, Stratified Log-rank Test — Stratified Log-rank Test P-value for Equality of Survival Curves; Hazard Ratio (HR) = 0.733, 95% CI 2-sided [0.364 to 1.479] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Mean Baseline and Unadjusted Mean Change From Baseline in Young-Mania Rating Scale (Y-MRS) Total Score Through Phase 2
Description: The Y-MRS consists of 11 items: 1) Elevated Mood, 2) Increased Motor Activity -Energy, 3) Sexual Interest, 4) Sleep, 5) Irritability, 6) Speech (Rate and Amount), 7) Language -Thought Disorder, 8) Content, 9) Disruptive-Aggressive Behavior, 10) Appearance, 11) Insight. Seven items are rated on a 0 to 4 scale, while 4 items (items 5, 6, 8 and 9) are rated on a 0 to 8 scale (twice the weight of the other items.) For all items, 0 is the "best" rating and 4 or 8 is the "worst" rating. Total Score is the sum of the ratings for all 11 items. The possible Total Scores are from 0 (best) to 60 (worst).
Time Frame: Baseline (end of ph 1), Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, and Phase 2 (Ph2) Endpoint. Phase 2 (13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout, + Confirmation of Partial Nonresponse Phase)
Population: Observed Cases (OC) data set; n=number of participants with measurement at given time point.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Lithium: Phase 2 (13 to 24 Week Stability and Maintenance of Stability Phase): aripiprazole 10-mg and 15-mg oral tablets and 250-mg and 300-mg oral lithium tablets
- Valproate: Phase 2 (13 to 24 Week Stability and Maintenance of Stability Phase): aripiprazole 10-mg and 15-mg oral tablets and 250-mg Depakote/valproic acid oral tablets
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 289 | 383
units on a scale
  Baseline (n=289, 383) | 23.15 (0.327) | 22.32 (0.252)
  Change from Baseline at Week 1 (n=277, 371) | -4.50 (0.312) | -4.86 (0.272)
  Change from Baseline at Week 2 (n=266, 355) | -7.90 (0.432) | -7.82 (0.351)
  Change from Baseline at Week 4 (n=245, 326) | -12.11 (0.454) | -10.75 (0.366)
  Change from Baseline at Week 6 (n=221, 305) | -13.92 (0.514) | -13.28 (0.394)
  Change from Baseline at Week 8 (n=201, 287) | -16.18 (0.495) | -14.84 (0.406)
  Change from Baseline at Week 12 (n=179, 253) | -17.74 (0.528) | -16.28 (0.427)
  Change from Baseline at Week 16 (n=138, 193) | -18.88 (0.639) | -17.55 (0.462)
  Change from Baseline at Week 20 (n=59, 99) | -20.37 (1.213) | -17.64 (0.741)
  Change from Baseline at Week 24 (n=22, 39) | -20.82 (1.550) | -19.77 (1.315)
  Change from Baseline at Ph2 endpoint (n=289, 383) | -14.78 (0.530) | -14.32 (0.429)

6. Secondary Outcome: Mean Baseline and Adjusted Mean Change From Baseline in Young-Mania Rating Scale (Y-MRS) Total Score Through Phase 3
Description: The Y-MRS consists of 11 items: 1) Elevated Mood, 2) Increased Motor Activity -Energy, 3) Sexual Interest, 4) Sleep, 5) Irritability, 6) Speech (Rate and Amount), 7) Language -Thought Disorder, 8) Content, 9) Disruptive-Aggressive Behavior, 10) Appearance, 11) Insight. 7 items are rated on a 0 to 4 scale, while 4 items (items 5, 6, 8 and 9) are rated on a 0 to 8 scale (twice the weight of the other items.) For all items, 0 is the "best" rating and 4 or 8 is the "worst" rating. Total Score is the sum of the ratings for all 11 items. The possible Total Scores are from 0 (best) to 60 (worst).
Time Frame: Baseline (end of Ph 2), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52 of Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: LOCF data set, phase 3 efficacy sample; n=number of participants with measurement at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Baseline (n=164, 162) | 4.03 (0.285) | 4.06 (0.280)
  Change at Week 4 (n=160, 162) | 0.47 (0.342) | 0.53 (0.332)
  Change at Week 8 (n=164, 162) | 0.91 (0.353) | 0.23 (0.346)
  Change at Week 12 (n=164, 162) | 1.53 (0.415) | 0.43 (0.408)
  Change at Week 16 (n=164, 162) | 1.74 (0.433) | 0.35 (0.425)
  Change at Week 20 (n=164, 162) | 2.29 (0.472) | 0.38 (0.463)
  Change at Week 24 (n=164, 162) | 2.42 (0.492) | 0.24 (0.483)
  Change at Week 28 (n=164, 162) | 3.02 (0.547) | 0.40 (0.537)
  Change at Week 32 (n=164, 162) | 2.72 (0.526) | 0.39 (0.516)
  Change at Week 36 (n=164, 162) | 3.04 (0.538) | 0.26 (0.528)
  Change at Week 40 (n=164, 162) | 2.82 (0.542) | 0.11 (0.532)
  Change at Week 44 (n=164, 162) | 3.19 (0.558) | 0.27 (0.548)
  Change at Week 48 (n=164, 162) | 3.15 (0.575) | 0.07 (0.564)
  Change at Week 52 (n=164, 162) | 2.93 (0.576) | -0.11 (0.565)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Baseline Comparison; Test type: Superiority or Other; p = 0.955, ANOVA/ANCOVA — Mean change from baseline: ANOVA model, controlling for treatment, mood stabilizer, index mood episode, and baseline value. Mean change from baseline: ANCOVA model, controlling for treatment, mood stabilizer, index mood episode, baseline value; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = 0.02, 95% CI 2-sided [-0.73 to 0.77]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 4 Comparison; Test type: Superiority or Other; p = 0.895, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = 0.06, 95% CI 2-sided [-0.83 to 0.95]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 8 Comparison; Test type: Superiority or Other; p = 0.144, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.69, 95% CI 2-sided [-1.61 to 0.24]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 12 Comparison; Test type: Superiority or Other; p = 0.047, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.10, 95% CI 2-sided [-2.19 to -0.01]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 16 Comparison; Test type: Superiority or Other; p = 0.017, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.39, 95% CI 2-sided [-2.52 to -0.25]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 20 Comparison; Test type: Superiority or Other; p = 0.003, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.91, 95% CI 2-sided [-3.15 to -0.68]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 24 Comparison; Test type: Superiority or Other; p < 0.001, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -2.18, 95% CI 2-sided [-3.47 to -0.89]
Statistical Analysis 8: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 28 Comparison; Test type: Superiority or Other; p < 0.001, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -2.62, 95% CI 2-sided [-4.06 to -1.19]
Statistical Analysis 9: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 32 Comparison; Test type: Superiority or Other; p < 0.001, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -2.33, 95% CI 2-sided [-3.70 to -0.95]
Statistical Analysis 10: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 36 Comparison; Test type: Superiority or Other; p < 0.001, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -2.78, 95% CI 2-sided [-4.19 to -1.37]
Statistical Analysis 11: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 40 Comparison; Test type: Superiority or Other; p < 0.001, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -2.71, 95% CI 2-sided [-4.13 to -1.29]
Statistical Analysis 12: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 44 Comparison; Test type: Superiority or Other; p < 0.001, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -2.92, 95% CI 2-sided [-4.38 to -1.46]
Statistical Analysis 13: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 48 Comparison; Test type: Superiority or Other; p < 0.001, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -3.08, 95% CI 2-sided [-4.59 to -1.57]
Statistical Analysis 14: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 52 Comparison; Test type: Superiority or Other; p < 0.001, ANOVA/ANCOVA — [p-value comment as in outcome 6, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -3.04, 95% CI 2-sided [-4.55 to -1.54]

7. Secondary Outcome: Mean Baseline and Unadjusted Mean Change From Baseline in Montgomery Åsberg Depression Rating Scale (MADRS) Total Score Through Phase 2 and at Phase 2 Endpoint
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. MADRS total score, a 10-item, ordinal rating scale (0=no symptoms; 60=most severe symptoms). Change from baseline=postbaseline score - baseline score. A negative change score indicates improvement.
Time Frame: Baseline (end of Ph 1), Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, and Phase 2 (Ph2) Endpoint. Phase 2 (13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout, and Confirmation of Partial Nonresponse Phase)
Population: Observed Cases (OC) data set; phase 2 endpoint was phase 2 efficacy sample. n=number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 289 | 383
units on a scale
  Mean Baseline (n=289, 383) | 10.97 (0.508) | 11.56 (0.432)
  Change from Baseline at Week 1 (n=277, 371) | -1.48 (0.295) | -1.51 (0.256)
  Change from Baseline at Week 2 (n=267, 355) | -2.23 (0.352) | -2.70 (0.329)
  Change from Baseline at Week 4 (n=245, 326) | -2.94 (0.391) | -3.16 (0.357)
  Change from Baseline at Week 6 (n=221, 305) | -2.92 (0.466) | -3.69 (0.383)
  Change from Baseline at Week 8 (n=201, 287) | -3.07 (0.460) | -3.64 (0.440)
  Change from Baseline at Week 12 (n=179, 253) | -2.82 (0.500) | -3.91 (0.398)
  Change from Baseline at Week 16 (n=138, 193) | -2.88 (0.698) | -4.28 (0.425)
  Change from Baseline at Week 20 (n=59, 99) | -4.68 (0.944) | -4.49 (0.676)
  Change from Baseline at Week 24 (n=22, 39) | -3.77 (1.298) | -5.15 (1.186)
  Change from Baseline at Ph2 Endpoint (n=289, 383) | -2.13 (0.461) | -2.54 (0.412)

8. Secondary Outcome: Mean Baseline and Adjusted Mean Change From Baseline in Montgomery Åsberg Depression Rating Scale (MADRS) Total Score Through Phase 3
Description: as for outcome 7
Time Frame: Baseline (end of Ph 2), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52. Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: LOCF data set, phase 3 efficacy sample; N=number of participants evaluated at time point; 4 participants in the Week 4 placebo group were not evaluated.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Mean Baseline (n=164, 162) | 4.41 (0.282) | 4.62 (0.277)
  Mean Change from Baseline at Week 4 (n=160, 162) | 1.92 (0.421) | 1.42 (0.411)
  Mean Change from Baseline at Week 8 (n=164, 162) | 2.27 (0.495) | 1.23 (0.488)
  Mean Change from Baseline at Week 12 (n=164, 162) | 2.42 (0.493) | 1.42 (0.486)
  Mean Change from Baseline at Week 16 (n=164, 162) | 2.12 (0.505) | 1.27 (0.498)
  Mean Change from Baseline at Week 20 (n=164, 162) | 2.61 (0.557) | 1.47 (0.549)
  Mean Change from Baseline at Week 24 (n=164, 162) | 2.92 (0.572) | 1.49 (0.564)
  Mean Change from Baseline at Week 28 (n=164, 162) | 3.14 (0.601) | 1.64 (0.594)
  Mean Change from Baseline at Week 32 (n=164, 162) | 3.32 (0.609) | 1.70 (0.601)
  Mean Change from Baseline at Week 36 (n=164, 162) | 3.03 (0.621) | 1.89 (0.612)
  Mean Change from Baseline at Week 40 (n=164, 162) | 3.18 (0.626) | 1.65 (0.618)
  Mean Change from Baseline at Week 44 (n=164, 162) | 3.10 (0.641) | 1.53 (0.632)
  Mean Change from Baseline at Week 48 (n=164, 162) | 3.57 (0.633) | 1.48 (0.624)
  Mean Change from Baseline at Week 52 (n=164, 162) | 3.47 (0.640) | 1.46 (0.632)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Baseline Comparison; Test type: Superiority or Other; p = 0.590, ANOVA/ANCOVA — Baseline: ANOVA model, controlling for treatment, mood stabilizer, and index mood episode. Mean change from baseline: ANCOVA model, controlling for treatment, mood stabilizer, index mood episode, baseline value; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = 0.20, 95% CI 2-sided [-0.54 to 0.94]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 4 Comparison; Test type: Superiority or Other; p = 0.371, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.50, 95% CI 2-sided [-1.59 to 0.60]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 8 Comparison; Test type: Superiority or Other; p = 0.113, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.04, 95% CI 2-sided [-2.33 to 0.25]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 12 Comparison; Test type: Superiority or Other; p = 0.128, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.00, 95% CI 2-sided [-2.28 to 0.29]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 16 Comparison; Test type: Superiority or Other; p = 0.205, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.85, 95% CI 2-sided [-2.16 to 0.47]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 20 Comparison; Test type: Superiority or Other; p = 0.125, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.13, 95% CI 2-sided [-2.59 to 0.32]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 24 Comparison; Test type: Superiority or Other; p = 0.061, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.43, 95% CI 2-sided [-2.92 to 0.06]
Statistical Analysis 8: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 28 Comparison; Test type: Superiority or Other; p = 0.060, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.51, 95% CI 2-sided [-3.07 to 0.06]
Statistical Analysis 9: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 32 Comparison; Test type: Superiority or Other; p = 0.046, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.62, 95% CI 2-sided [-3.21 to -0.03]
Statistical Analysis 10: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 36 Comparison; Test type: Superiority or Other; p = 0.164, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.15, 95% CI 2-sided [-2.77 to 0.47]
Statistical Analysis 11: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 40 Comparison; Test type: Superiority or Other; p = 0.066, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.53, 95% CI 2-sided [-3.16 to 0.10]
Statistical Analysis 12: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 44 Comparison; Test type: Superiority or Other; p = 0.066, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -1.57, 95% CI 2-sided [-3.24 to 0.10]
Statistical Analysis 13: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 48 Comparison; Test type: Superiority or Other; p = 0.014, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -2.08, 95% CI 2-sided [-3.73 to -0.43]
Statistical Analysis 14: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 52 Comparison; Test type: Superiority or Other; p = 0.019, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -2.01, 95% CI 2-sided [-3.68 to -0.34]

9. Secondary Outcome: Unadjusted Mean Change Baseline and Mean Change From Baseline in the CGI-BP Severity of Illness (Overall) Through Phase 2
Description: as for outcome 2
Time Frame: Baseline (end of Ph 1), Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, and Phase 2 Endpoint. Phase 2 (13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout, and Confirmation of Partial Nonresponse Phase)
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 289 | 383
units on a scale
  Mean Baseline (BL) (n=289, 383) | 4.25 (0.040) | 4.08 (0.036)
  Mean Change from BL to Week 1 (n=275, 370) | -0.52 (0.046) | -0.53 (0.040)
  Mean Change from BL to Week 2 (n=267, 354) | -1.05 (0.061) | -0.97 (0.054)
  Mean Change from BL to Week 4 (n=245, 326) | -1.56 (0.074) | -1.31 (0.059)
  Mean Change from BL to Week 6 (n=219, 305) | -1.86 (0.084) | -1.62 (0.063)
  Mean Change from BL to Week 8 (n=200, 287) | -2.17 (0.081) | -1.80 (0.069)
  Mean Change from BL to Week 12 (n=179, 252) | -2.31 (0.097) | -1.99 (0.078)
  Mean Change from BL to Week 16 (n=138, 193) | -2.57 (0.106) | -2.17 (0.079)
  Mean Change from BL to Week 20 (n=59, 99) | -2.71 (0.181) | -2.14 (0.118)
  Mean Change from BL to Week 24 (n=22, 39) | -2.73 (0.220) | -2.38 (0.186)
  Mean Change from BL to Phase 2 Endpoint(n=289,383) | -1.90 (0.085) | -1.66 (0.070)

10. Secondary Outcome: Baseline and Adjusted Mean Change From Baseline in the CGI-BP Severity of Illness (Overall) Through Phase 3
Description: as for outcome 2
Time Frame: as for outcome 8
Population: LOCF data set, phase 3 efficacy sample; 4 participants in the Week 4 placebo group were not evaluated.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Mean Baseline | 1.65 (0.065) | 1.70 (0.064)
  Mean Change from Baseline At Week 4 (n=160, 162) | 0.25 (0.072) | 0.27 (0.070)
  Mean Change from Baseline At Week 8 | 0.32 (0.080) | 0.21 (0.079)
  Mean Change from Baseline At Week 12 | 0.40 (0.087) | 0.26 (0.085)
  Mean Change from Baseline At Week 16 | 0.44 (0.088) | 0.26 (0.087)
  Mean Change from Baseline At Week 20 | 0.51 (0.095) | 0.29 (0.094)
  Mean Change from Baseline At Week 24 | 0.56 (0.097) | 0.25 (0.095)
  Mean Change from Baseline At Week 28 | 0.62 (0.101) | 0.32 (0.099)
  Mean Change from Baseline At Week 32 | 0.61 (0.102) | 0.30 (0.100)
  Mean Change from Baseline At Week 36 | 0.62 (0.103) | 0.33 (0.101)
  Mean Change from Baseline At Week 40 | 0.57 (0.104) | 0.28 (0.102)
  Mean Change from Baseline At Week 44 | 0.64 (0.105) | 0.30 (0.103)
  Mean Change from Baseline At Week 48 | 0.68 (0.106) | 0.28 (0.104)
  Mean Change from Baseline At Week 52 | 0.66 (0.106) | 0.31 (0.104)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Baseline Comparison; Test type: Superiority or Other; p = 0.597, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = 0.05, 95% CI 2-sided [-0.13 to 0.22]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 4 Comparison; Test type: Superiority or Other; p = 0.838, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = 0.02, 95% CI 2-sided [-0.17 to 0.21]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 8 Comparison; Test type: Superiority or Other; p = 0.291, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.11, 95% CI 2-sided [-0.32 to 0.10]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 12 Comparison; Test type: Superiority or Other; p = 0.219, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.14, 95% CI 2-sided [-0.37 to 0.08]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 16 Comparison; Test type: Superiority or Other; p = 0.133, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.18, 95% CI 2-sided [-0.41 to 0.05]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 20 Comparison; Test type: Superiority or Other; p = 0.092, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.21, 95% CI 2-sided [-0.46 to 0.04]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 24 Comparison; Test type: Superiority or Other; p = 0.018, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.31, 95% CI 2-sided [-0.56 to -0.05]
Statistical Analysis 8: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 28 Comparison; Test type: Superiority or Other; p = 0.029, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.29, 95% CI 2-sided [-0.56 to -0.03]
Statistical Analysis 9: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 32 Comparison; Test type: Superiority or Other; p = 0.024, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.31, 95% CI 2-sided [-0.57 to -0.04]
Statistical Analysis 10: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 36 Comparison; Test type: Superiority or Other; p = 0.035, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.29, 95% CI 2-sided [-0.56 to -0.02]
Statistical Analysis 11: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 40 Comparison; Test type: Superiority or Other; p = 0.038, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.29, 95% CI 2-sided [-0.56 to -0.02]
Statistical Analysis 12: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 44 Comparison; Test type: Superiority or Other; p = 0.015, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.34, 95% CI 2-sided [-0.62 to -0.07]
Statistical Analysis 13: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 48 Comparison; Test type: Superiority or Other; p = 0.006, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.39, 95% CI 2-sided [-0.67 to -0.12]
Statistical Analysis 14: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 52 Comparison; Test type: Superiority or Other; p = 0.015, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.35, 95% CI 2-sided [-0.62 to -0.07]

11. Secondary Outcome: Unadjusted Mean Change Baseline and Mean Change From Baseline in the CGI-BP Severity of Illness (Depression) Through Phase 2
Description: Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change in patients with bipolar disorder. Patients are rated on Change from baseline (mania, depression and overall bipolar illness) items (also a 7-point scale [1 to 7], with 1 being normal and 7 being very severely ill). A negative change score signifies improvement.
Time Frame: Baseline (end of Ph 1), Weeks 1, 2, 4,6, 8, 12, 16, 20, 24, and Phase 2 Endpoint. Phase 2 (13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout, and Confirmation of Partial Nonresponse Phase)
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 289 | 383
units on a scale
  Mean Baseline (BL) (n=289, 383) | 2.16 (0.076) | 2.33 (0.069)
  Mean Change from BL to Week 1 (n=275, 370) | -0.16 (0.041) | -0.19 (0.040)
  Mean Change from BL to Week 2 (n=267, 354) | -0.22 (0.053) | -0.33 (0.050)
  Mean Change from BL to Week 4 (n=245, 326) | -0.29 (0.058) | -0.39 (0.055)
  Mean Change from BL to Week 6 (n=219, 305) | -0.31 (0.068) | -0.43 (0.061)
  Mean Change from BL to Week 8 (n=200, 287) | -0.30 (0.077) | -0.37 (0.066)
  Mean Change from BL to Week 12 (n=179, 252) | -0.17 (0.077) | -0.35 (0.069)
  Mean Change from BL to Week 16 (n=138, 193) | -0.21 (0.109) | -0.36 (0.078)
  Mean Change from BL to Week 20 (n=59, 99) | -0.27 (0.149) | -0.37 (0.116)
  Mean Change from BL to Week 24 (n=22, 39) | -0.23 (0.227) | -0.46 (0.217)
  Mean Change from BL to Phase 2 Endpoint(n=289,383) | -0.16 (0.069) | -0.26 (0.063)

12. Secondary Outcome: Baseline and Adjusted Mean Change From Baseline in CGI-BP Severity of Illness (Depression) Score Through Phase 3
Description: as for outcome 2
Time Frame: as for outcome 8
Population: LOCF data set, phase 3 efficacy sample; 4 participants in the Week 4 placebo group were not evaluated.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Baseline Mean | 1.43 (0.049) | 1.47 (0.048)
  Mean Change from Baseline at Week 4 (n=160, 162) | 0.30 (0.067) | 0.29 (0.065)
  Mean Change from Baseline at Week 8 | 0.35 (0.073) | 0.24 (0.072)
  Mean Change from Baseline at Week 12 | 0.37 (0.077) | 0.23 (0.076)
  Mean Change from Baseline at Week 16 | 0.35 (0.078) | 0.24 (0.077)
  Mean Change from Baseline at Week 20 | 0.41 (0.084) | 0.28 (0.083)
  Mean Change from Baseline at Week 24 | 0.44 (0.086) | 0.27 (0.085)
  Mean Change from Baseline at Week 28 | 0.50 (0.091) | 0.28 (0.090)
  Mean Change from Baseline at Week 32 | 0.53 (0.092) | 0.27 (0.091)
  Mean Change from Baseline at Week 36 | 0.49 (0.092) | 0.32 (0.091)
  Mean Change from Baseline at Week 40 | 0.47 (0.093) | 0.28 (0.091)
  Mean Change from Baseline at Week 44 | 0.46 (0.094) | 0.28 (0.093)
  Mean Change from Baseline at Week 48 | 0.50 (0.094) | 0.27 (0.092)
  Mean Change from Baseline at Week 52 | 0.51 (0.094) | 0.30 (0.093)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Baseline Comparison; Test type: Superiority or Other; p = 0.588, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = 0.04, 95% CI 2-sided [-0.09 to 0.16]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 4 Comparison; Test type: Superiority or Other; p = 0.922, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.01, 95% CI 2-sided [-0.18 to 0.16]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 8 Comparison; Test type: Superiority or Other; p = 0.266, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.11, 95% CI 2-sided [-0.30 to 0.08]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 12 Comparison; Test type: Superiority or Other; p = 0.159, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.14, 95% CI 2-sided [-0.34 to 0.06]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 16 Comparison; Test type: Superiority or Other; p = 0.305, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.11, 95% CI 2-sided [-0.31 to 0.10]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 20 Comparison; Test type: Superiority or Other; p = 0.251, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.13, 95% CI 2-sided [-0.35 to 0.09]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 24 Comparison; Test type: Superiority or Other; p = 0.135, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.17, 95% CI 2-sided [-0.40 to 0.05]
Statistical Analysis 8: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 28 Comparison; Test type: Superiority or Other; p = 0.073, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.22, 95% CI 2-sided [-0.46 to 0.02]
Statistical Analysis 9: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 32 Comparison; Test type: Superiority or Other; p = 0.034, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.26, 95% CI 2-sided [-0.50 to -0.02]
Statistical Analysis 10: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 36 Comparison; Test type: Superiority or Other; p = 0.174, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.17, 95% CI 2-sided [-0.41 to 0.07]
Statistical Analysis 11: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 40 Comparison; Test type: Superiority or Other; p = 0.132, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.19, 95% CI 2-sided [-0.43 to 0.06]
Statistical Analysis 12: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 44 Comparison; Test type: Superiority or Other; p = 0.152, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.18, 95% CI 2-sided [-0.42 to 0.07]
Statistical Analysis 13: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 48 Comparison; Test type: Superiority or Other; p = 0.060, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.23, 95% CI 2-sided [-0.48 to 0.01]
Statistical Analysis 14: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 52 Comparison; Test type: Superiority or Other; p = 0.085, ANOVA/ANCOVA — [p-value comment as in outcome 8, analysis 1]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.22, 95% CI 2-sided [-0.46 to 0.03]

13. Secondary Outcome: Unadjusted Mean Change From Preceding Phase in the CGI-BP (Mania) Through Phase 2
Description: Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change from baseline in patients with bipolar disorder. Patients are rated on mania, depression and overall change from preceding phase items on a 7-point scale [1 to 7], with 1 being very much improved and 7 being very much worse).
Time Frame: Weeks 1, 2, 4,6, 8, 12, 16, 20, 24, and Phase 2 Endpoint. Phase 2 (13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout, and Confirmation of Partial Nonresponse Phase)
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 289 | 382
units on a scale
  Mean Change from BL to Week 1 (n=274, 369) | 3.15 (0.055) | 3.09 (0.049)
  Mean Change from BL to Week 2 (n=265, 353) | 2.61 (0.062) | 2.58 (0.054)
  Mean Change from BL to Week 4 (n=245, 325) | 2.14 (0.060) | 2.24 (0.056)
  Mean Change from BL to Week 6 (n=219, 305) | 1.95 (0.065) | 1.97 (0.056)
  Mean Change from BL to Week 8 (n=200, 287) | 1.73 (0.062) | 1.80 (0.055)
  Mean Change from BL to Week 12 (n=179, 252) | 1.66 (0.074) | 1.65 (0.053)
  Mean Change from BL to Week 16 (n=138, 193) | 1.54 (0.082) | 1.61 (0.056)
  Mean Change from BL to Week 20 (n=59, 99) | 1.69 (0.161) | 1.68 (0.087)
  Mean Change from BL to Week 24 (n=22, 39) | 1.64 (0.214) | 1.67 (0.181)
  Mean Change from BL to Phase 2 Endpoint(n=289,382) | 1.95 (0.071) | 1.94 (0.056)

14. Secondary Outcome: Unadjusted Mean Baseline and Mean Change From Baseline in the CGI-BP Severity of Illness (Mania) Through Phase 2
Description: as for outcome 11
Time Frame: as for outcome 11
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 289 | 383
units on a scale
  Mean Baseline (BL) (n=289, 383) | 4.22 (0.040) | 4.06 (0.035)
  Mean Change from BL to Week 1 (n=275, 370) | -0.58 (0.047) | -0.58 (0.042)
  Mean Change from BL to Week 2 (n=267, 354) | -1.15 (0.064) | -1.06 (0.055)
  Mean Change from BL to Week 4 (n=245, 326) | -1.73 (0.075) | -1.45 (0.062)
  Mean Change from BL to Week 6 (n=219, 305) | -2.04 (0.081) | -1.82 (0.065)
  Mean Change from BL to Week 8 (n=200, 287) | -2.40 (0.076) | -2.06 (0.067)
  Mean Change from BL to Week 12 (n=179, 252) | -2.60 (0.081) | -2.27 (0.071)
  Mean Change from BL to Week 16 (n=138, 193) | -2.83 (0.086) | -2.40 (0.075)
  Mean Change from BL to Week 20 (n=59, 99) | -2.93 (0.162) | -2.32 (0.115)
  Mean Change from BL to Week 24 (n=22, 39) | -2.91 (0.185) | -2.56 (0.163)
  Mean Change from BL to Phase 2 Endpoint(n=289,383) | -2.21 (0.079) | -2.01 (0.066)

15. Secondary Outcome: Adjusted Mean Change in CGI-BP From Preceding Phase (Mania) Through Phase 3
Description: as for outcome 2
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52. Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: LOCF data set, phase 3 efficacy sample; 4 participants in the Week 4 placebo group were not evaluated.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Mean Change at Week 4 (n=160, 162) | 2.96 (0.111) | 3.00 (0.108)
  Mean Change at Week 8 | 3.17 (0.113) | 2.98 (0.111)
  Mean Change at Week 12 | 3.14 (0.118) | 3.03 (0.116)
  Mean Change at Week 16 | 3.27 (0.118) | 2.98 (0.115)
  Mean Change at Week 20 | 3.29 (0.120) | 3.03 (0.118)
  Mean Change at Week 24 | 3.26 (0.125) | 2.96 (0.123)
  Mean Change at Week 28 | 3.37 (0.126) | 3.01 (0.124)
  Mean Change at Week 32 | 3.31 (0.124) | 3.00 (0.122)
  Mean Change at Week 36 | 3.37 (0.125) | 2.94 (0.123)
  Mean Change at Week 40 | 3.32 (0.126) | 2.94 (0.124)
  Mean Change at Week 44 | 3.33 (0.128) | 2.96 (0.125)
  Mean Change at Week 48 | 3.35 (0.130) | 2.96 (0.128)
  Mean Change at Week 52 | 3.29 (0.131) | 2.89 (0.129)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 4 Comparison; Test type: Superiority or Other; p = 0.774, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = 0.04, 95% CI 2-sided [-0.25 to 0.33]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 8 Comparison; Test type: Superiority or Other; p = 0.213, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.19, 95% CI 2-sided [-0.49 to 0.11]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 12 Comparison; Test type: Superiority or Other; p = 0.465, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.12, 95% CI 2-sided [-0.43 to 0.20]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 16 Comparison; Test type: Superiority or Other; p = 0.068, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.29, 95% CI 2-sided [-0.59 to 0.02]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 20 Comparison; Test type: Superiority or Other; p = 0.095, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.27, 95% CI 2-sided [-0.58 to 0.05]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 24 Comparison; Test type: Superiority or Other; p = 0.082, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.29, 95% CI 2-sided [-0.62 to 0.04]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 28 Comparison; Test type: Superiority or Other; p = 0.033, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.36, 95% CI 2-sided [-0.69 to -0.03]
Statistical Analysis 8: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 32 Comparison; Test type: Superiority or Other; p = 0.062, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.31, 95% CI 2-sided [-0.64 to 0.02]
Statistical Analysis 9: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 36 Comparison; Test type: Superiority or Other; p = 0.011, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.43, 95% CI 2-sided [-0.76 to -0.10]
Statistical Analysis 10: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 40 Comparison; Test type: Superiority or Other; p = 0.027, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.37, 95% CI 2-sided [-0.70 to -0.04]
Statistical Analysis 11: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 44 Comparison; Test type: Superiority or Other; p = 0.029, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.37, 95% CI 2-sided [-0.71 to -0.04]
Statistical Analysis 12: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 48 Comparison; Test type: Superiority or Other; p = 0.022, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.40, 95% CI 2-sided [-0.74 to -0.06]
Statistical Analysis 13: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 52 Comparison; Test type: Superiority or Other; p = 0.023, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.40, 95% CI 2-sided [-0.75 to -0.06]

16. Secondary Outcome: Unadjusted Mean Change From Preceding Phase in the CGI-BP (Depression) Through Phase 2
Description: Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change in patients with bipolar disorder. Patients are rated on Change from Preceding Phase (mania, depression and overall bipolar illness) items (also a 7-point scale [1 to 7], with 1 being very much improved and 7 being very much worse).
Time Frame: Weeks 1, 2, 4, 6, 8, 12, 16, 20, 24, and Phase 2 Endpoint. Phase 2 (13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout, and Confirmation of Partial Nonresponse Phase)
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 289 | 382
units on a scale
  Mean Change from BL to Week 1 (n=274, 368) | 3.56 (0.054) | 3.40 (0.057)
  Mean Change from BL to Week 2 (n=265, 353) | 3.42 (0.061) | 3.25 (0.066)
  Mean Change from BL to Week 4 (n=245, 325) | 3.35 (0.074) | 3.19 (0.071)
  Mean Change from BL to Week 6 (n=219, 305) | 3.22 (0.083) | 3.13 (0.078)
  Mean Change from BL to Week 8 (n=200, 287) | 3.13 (0.090) | 3.11 (0.084)
  Mean Change from BL to Week 12 (n=179, 250) | 3.28 (0.094) | 3.06 (0.087)
  Mean Change from BL to Week 16 (n=138, 193) | 3.30 (0.117) | 2.99 (0.100)
  Mean Change from BL to Week 20 (n=59, 99) | 3.24 (0.173) | 3.18 (0.129)
  Mean Change from BL to Week 24 (n=22, 39) | 2.91 (0.278) | 3.15 (0.251)
  Mean Change from BL to Phase 2 Endpoint(n=289,382) | 3.30 (0.080) | 3.26 (0.075)

17. Secondary Outcome: Adjusted Mean Change in CGI-BP From Preceding Phase (Depression) Through Phase 3
Description: Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change from baseline (in this case, preceding phase) in patients with bipolar disorder. Patients are rated on mania, depression and overall bipolar illness items on a 7-point scale [1 to 7], with 1 being very much improved and 7 being very much worse).
Time Frame: as for outcome 15
Population: LOCF data set, phase 3 efficacy sample; 4 participants in the Week 4 placebo group were not evaluated.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Mean Change at Week 4 (n=160, 162) | 3.46 (0.102) | 3.56 (0.100)
  Mean Change at Week 8 | 3.55 (0.103) | 3.52 (0.101)
  Mean Change at Week 12 | 3.51 (0.106) | 3.45 (0.104)
  Mean Change at Week 16 | 3.52 (0.108) | 3.45 (0.107)
  Mean Change at Week 20 | 3.58 (0.111) | 3.53 (0.109)
  Mean Change at Week 24 | 3.63 (0.112) | 3.54 (0.110)
  Mean Change at Week 28 | 3.65 (0.116) | 3.52 (0.114)
  Mean Change at Week 32 | 3.69 (0.116) | 3.49 (0.114)
  Mean Change at Week 36 | 3.62 (0.119) | 3.52 (0.117)
  Mean Change at Week 40 | 3.55 (0.120) | 3.47 (0.118)
  Mean Change at Week 44 | 3.52 (0.121) | 3.49 (0.120)
  Mean Change at Week 48 | 3.58 (0.121) | 3.44 (0.120)
  Mean Change at Week 52 | 3.56 (0.122) | 3.44 (0.120)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 4 Comparison; Test type: Superiority or Other; p = 0.486, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = 0.09, 95% CI 2-sided [-0.17 to 0.36]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 8 Comparison; Test type: Superiority or Other; p = 0.793, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.04, 95% CI 2-sided [-0.30 to 0.23]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 12 Comparison; Test type: Superiority or Other; p = 0.665, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.06, 95% CI 2-sided [-0.34 to 0.22]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 16 Comparison; Test type: Superiority or Other; p = 0.650, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.07, 95% CI 2-sided [-0.35 to 0.22]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 20 Comparison; Test type: Superiority or Other; p = 0.705, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.06, 95% CI 2-sided [-0.34 to 0.23]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 24 Comparison; Test type: Superiority or Other; p = 0.572, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.08, 95% CI 2-sided [-0.38 to 0.21]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 28 Comparison; Test type: Superiority or Other; p = 0.418, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.12, 95% CI 2-sided [-0.43 to 0.18]
Statistical Analysis 8: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 32 Comparison; Test type: Superiority or Other; p = 0.185, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.20, 95% CI 2-sided [-0.51 to 0.10]
Statistical Analysis 9: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 36 Comparison; Test type: Superiority or Other; p = 0.536, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.10, 95% CI 2-sided [-0.41 to 0.21]
Statistical Analysis 10: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 40 Comparison; Test type: Superiority or Other; p = 0.637, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.07, 95% CI 2-sided [-0.39 to 0.24]
Statistical Analysis 11: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 44 Comparison; Test type: Superiority or Other; p = 0.875, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.03, 95% CI 2-sided [-0.34 to 0.29]
Statistical Analysis 12: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 48 Comparison; Test type: Superiority or Other; p = 0.378, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.14, 95% CI 2-sided [-0.46 to 0.17]
Statistical Analysis 13: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 52 Comparison; Test type: Superiority or Other; p = 0.474, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.12, 95% CI 2-sided [-0.43 to 0.20]

18. Secondary Outcome: Unadjusted Mean Change From Preceding Phase in the CGI-BP (Overall) Through Phase 2
Description: as for outcome 17
Time Frame: as for outcome 16
Population: as for outcome 7
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 289 | 382
units on a scale
  Mean Change from BL to Week 1 (n=274, 369) | 3.20 (0.054) | 3.13 (0.048)
  Mean Change from BL to Week 2 (n=265, 353) | 2.70 (0.063) | 2.69 (0.057)
  Mean Change from BL to Week 4 (n=245, 325) | 2.27 (0.063) | 2.40 (0.060)
  Mean Change from BL to Week 6 (n=219, 305) | 2.11 (0.069) | 2.19 (0.064)
  Mean Change from BL to Week 8 (n=200, 287) | 1.94 (0.073) | 2.08 (0.070)
  Mean Change from BL to Week 12 (n=179, 252) | 1.87 (0.081) | 1.94 (0.071)
  Mean Change from BL to Week 16 (n=138, 193) | 1.74 (0.096) | 1.80 (0.069)
  Mean Change from BL to Week 20 (n=59, 99) | 1.81 (0.156) | 1.90 (0.112)
  Mean Change from BL to Week 24 (n=22, 39) | 1.68 (0.212) | 1.82 (0.226)
  Mean Change from BL to Phase 2 Endpoint(n=289,382) | 2.26 (0.082) | 2.37 (0.072)

19. Secondary Outcome: Adjusted Mean Change in CGI-BP From Preceding Phase (Overall) Through Phase 3
Description: as for outcome 17
Time Frame: as for outcome 15
Population: LOCF data set, phase 3 efficacy sample; 4 participants in the Week 4 placebo group were not evaluated.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Mean Change at Week 4 (n=160, 162) | 3.17 (0.113) | 3.27 (0.110)
  Mean Change at Week 8 | 3.36 (0.118) | 3.22 (0.116)
  Mean Change at Week 12 | 3.34 (0.122) | 3.27 (0.120)
  Mean Change at Week 16 | 3.45 (0.121) | 3.22 (0.119)
  Mean Change at Week 20 | 3.53 (0.125) | 3.31 (0.122)
  Mean Change at Week 24 | 3.60 (0.127) | 3.31 (0.125)
  Mean Change at Week 28 | 3.65 (0.130) | 3.31 (0.127)
  Mean Change at Week 32 | 3.63 (0.130) | 3.29 (0.128)
  Mean Change at Week 36 | 3.61 (0.132) | 3.28 (0.130)
  Mean Change at Week 40 | 3.54 (0.133) | 3.24 (0.131)
  Mean Change at Week 44 | 3.57 (0.135) | 3.28 (0.132)
  Mean Change at Week 48 | 3.63 (0.136) | 3.26 (0.134)
  Mean Change at Week 52 | 3.58 (0.138) | 3.25 (0.135)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 4 Comparison; Test type: Superiority or Other; p = 0.488, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = 0.10, 95% CI 2-sided [-0.19 to 0.40]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 8 Comparison; Test type: Superiority or Other; p = 0.349, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.15, 95% CI 2-sided [-0.46 to 0.16]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 12 Comparison; Test type: Superiority or Other; p = 0.653, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.07, 95% CI 2-sided [-0.39 to 0.25]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 16 Comparison; Test type: Superiority or Other; p = 0.141, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.24, 95% CI 2-sided [-0.56 to 0.08]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 20 Comparison; Test type: Superiority or Other; p = 0.196, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.22, 95% CI 2-sided [-0.54 to 0.11]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 24 Comparison; Test type: Superiority or Other; p = 0.088, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.29, 95% CI 2-sided [-0.62 to 0.04]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 28 Comparison; Test type: Superiority or Other; p = 0.047, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.34, 95% CI 2-sided [-0.68 to -0.01]
Statistical Analysis 8: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 32 Comparison; Test type: Superiority or Other; p = 0.057, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.33, 95% CI 2-sided [-0.67 to 0.01]
Statistical Analysis 9: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 36 Comparison; Test type: Superiority or Other; p = 0.063, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.33, 95% CI 2-sided [-0.68 to 0.02]
Statistical Analysis 10: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 40 Comparison; Test type: Superiority or Other; p = 0.091, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.30, 95% CI 2-sided [-0.65 to 0.05]
Statistical Analysis 11: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 44 Comparison; Test type: Superiority or Other; p = 0.105, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.29, 95% CI 2-sided [-0.64 to 0.06]
Statistical Analysis 12: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 48 Comparison; Test type: Superiority or Other; p = 0.047, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.36, 95% CI 2-sided [-0.72 to -0.01]
Statistical Analysis 13: Comparison: Placebo vs Aripiprazole; Aripiprazole - Placebo; Week 52 Comparison; Test type: Superiority or Other; p = 0.073, ANOVA/ANCOVA — [p-value comment as in outcome 2, analysis 2]; Means, differences in means, 95% CI for the differences, and p-values are based on the ANOVA/ANCOVA model; Difference = -0.33, 95% CI 2-sided [-0.69 to 0.03]

20. Secondary Outcome: Number of Participants Maintaining Remission During Phase 3
Description: Remission is defined as Y-MRS Total Score <=12 and MADRS Total Score <=12.
Time Frame: as for outcome 15
Population: Observed cases data set, Phase 3 Efficacy Sample
Measure: Number; unit: participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 160 | 162
participants
  Week 4 (n=160, 162) | 142 | 142
  Week 8 (n=152, 145) | 138 | 136
  Week 12 (n=144, 136) | 133 | 126
  Week 16 (n=138, 131) | 122 | 126
  Week 20 (n=131, 127) | 115 | 117
  Week 24 (n=115, 122) | 107 | 119
  Week 28 (n=114, 122) | 100 | 115
  Week 32 (n=104, 119) | 99 | 112
  Week 36 (n=99, 108) | 91 | 104
  Week 40 (n=100, 110) | 93 | 109
  Week 44 (n=91, 109) | 81 | 102
  Week 48 (n=92, 102) | 85 | 101
  Week 52 (n=89, 97) | 82 | 95
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Week 4; Test type: Superiority or Other; p = 0.910, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.00, 95% CI 2-sided [0.92 to 1.08] — Aripiprazole/Placebo
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 8; Test type: Superiority or Other; p = 0.300, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.04, 95% CI 2-sided [0.97 to 1.11] — Aripiprazole/Placebo
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Week 12; Test type: Superiority or Other; p = 0.744, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.01, 95% CI 2-sided [0.95 to 1.08] — Aripiprazole/Placebo
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Week 16; Test type: Superiority or Other; p = 0.015, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.09, 95% CI 2-sided [1.02 to 1.17] — Aripiprazole/Placebo
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Week 20; Test type: Superiority or Other; p = 0.264, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.05, 95% CI 2-sided [0.97 to 1.14] — Aripiprazole/Placebo
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Week 24; Test type: Superiority or Other; p = 0.090, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.05, 95% CI 2-sided [0.99 to 1.11] — Aripiprazole/Placebo
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Week 28; Test type: Superiority or Other; p = 0.056, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.08, 95% CI 2-sided [1.00 to 1.17] — Aripiprazole/Placebo
Statistical Analysis 8: Comparison: Placebo vs Aripiprazole; Week 32; Test type: Superiority or Other; p = 0.756, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 0.99, 95% CI 2-sided [0.93 to 1.05] — Aripiprazole/Placebo
Statistical Analysis 9: Comparison: Placebo vs Aripiprazole; Week 36; Test type: Superiority or Other; p = 0.177, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.05, 95% CI 2-sided [0.98 to 1.13] — Aripiprazole/Placebo
Statistical Analysis 10: Comparison: Placebo vs Aripiprazole; Week 40; Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.07, 95% CI 2-sided [1.01 to 1.13] — Aripiprazole/Placebo
Statistical Analysis 11: Comparison: Placebo vs Aripiprazole; Week 44; Test type: Superiority or Other; p = 0.216, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.06, 95% CI 2-sided [0.96 to 1.16] — Aripiprazole/Placebo
Statistical Analysis 12: Comparison: Placebo vs Aripiprazole; Week 48; Test type: Superiority or Other; p = 0.017, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.07, 95% CI 2-sided [1.01 to 1.15] — Aripiprazole/Placebo
Statistical Analysis 13: Comparison: Placebo vs Aripiprazole; Week 52; Test type: Superiority or Other; p = 0.083, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel General Association Test controlling for mood stabilizer and index mood episode; Ratio of Remission Rate = 1.06, 95% CI 2-sided [0.99 to 1.13] — Aripiprazole/Placebo

21. Secondary Outcome: Proportion of Participants Discontinuing For Any Reason Through Week 52 (During Phase 3)
Time Frame: Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: Randomized Sample
Measure: Number; unit: Proportion of Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 169 | 168
Proportion of Participants | 0.473 | 0.387
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Test type: Superiority or Other; p = 0.132, Stratified Log Rank Test; Stratified Log Rank Test p-value for equality of survival curves; Cox Proportional Hazard = 0.78, 95% CI 2-sided [0.56 to 1.08]

22. Secondary Outcome: Deaths, Serious Adverse Events (SAEs), Adverse Events (AEs), and Discontinuations Due to AEs During Phase 2
Description: Participants with Adverse Events (AEs), Deaths, Serious AEs (SAEs), and AEs leading to study discontinuation. AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition. SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a cancer, is a congenital anomaly/birth defect, results in the development of drug dependency or drug abuse, is an important medical event.
Time Frame: During Phase 2 (a 13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout and Confirmation of Partial Nonresponse Phase)
Population: Phase 2 Safety Sample
Measure: Number; unit: Participants
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 292 | 390
Participants
  Deaths | 0 | 0
  SAEs | 5 | 10
  Discontinuations due to AEs | 38 | 50
  Any AE | 226 | 287
  Treatment-related AEs in >=2% of Participants | 188 | 233
  Any Extrapyramidal Syndrome-Related AE | 108 | 113

23. Secondary Outcome: Treatment-Emergent Adverse Events in >=5 Percent of Participants, by Severity, During Phase 2
Description: AE is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition. By Common Terminology Criteria Version 3.0 (CTC v3) Grade (Gr): Gr 1 (mild); Gr 2 (moderate); Gr 3 (severe); Gr 4 (life-threatening); Gr 5 (death).
Time Frame: During Phase 2. Phase 2 (13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout, and Confirmation of Partial Nonresponse Phase)
Population: Phase 2 Safety Sample
Measure: Number; unit: Participants
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 292 | 390
Participants
  Any Adverse Event | 226 | 287
  Mild/Grade 1 | 172 | 219
  Moderate/Grade 2 | 109 | 165
  Severe/Grade 3 | 20 | 31
  Very Severe/Grade 4 | 2 | 1

24. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Electrocardiogram (ECG) Abnormalities During Phase 2
Description: Sinus Tachycardia: ≥120bpm+↑≥15bpm+no current diagnosis of supraventricular (SV) or ventricular tachycardia or atrial fibrillation (AF) or flutter or other rhythm abnormality (RA). Sinus Bradycardia:≥50bpm+↓≥15bpm+no current diagnosis of AF or flutter or other RA. AF:not present→present or present at rate <100bpm pretreatment to present with rate ≥100bpm+increase of ≥15bpm. AV=atrioventricular; PR=PR interval. Other Intraventricular Block: QRS wave ≥0.12 sec+↑≥0.02 sec+no current diagnosis of left or right bundle branch block. Old Infarction not present→present at ≥12 weeks post study entry.
Time Frame: Phase 2 (a 13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout and Confirmation of Partial Nonresponse Phase)
Population: Phase 2 Safety Sample
Measure: Number; unit: Participants
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 292 | 390
Participants
  Tachycardia ≥ 120 bpm and ↑ ≥ 15 bpm | 0 | 2
  Bradycardia ≤ 50 bpm and ↓ 15 bpm | 0 | 4
  Sinus Tachycardia (see description) | 0 | 2
  Sinus Bradycardia (see description) | 0 | 4
  SV Premature Beat - not present → present | 2 | 2
  Ventricular Premature Beat - not present → present | 2 | 1
  SV Tachycardia not present → present | 0 | 0
  Ventricular Tachycardia not present → present | 0 | 0
  Atrial Fibrillation (see description) | 0 | 0
  Atrial Flutter not present → present | 0 | 0
  1st Degree AV Block PR ≥0.20 sec and ↑ ≥0.05 sec | 0 | 0
  2nd Degree AV Block not present → present | 0 | 0
  3rd Degree AV Block not present → present | 0 | 0
  Left Bundle Branch Block not present → present | 11 | 7
  Right Bundle Branch Block not present → present | 5 | 2
  Pre-excitation Syndrome not present → present | 0 | 0
  Other Intraventricular Block (see description) | 0 | 0
  Acute Infarction not present → present | 1 | 0
  Subacute (Recent) Infarction not present → present | 1 | 1
  Old Infarction not present → present at >=12 weeks | 0 | 0
  Myocardial Ischemia not present → present | 0 | 0
  Symmetrical T-Wave Inversion not present → present | 1 | 0
  QTc Bazett (QTcB) > 450 msec | 15 | 8
  QTc Frederica (QTcF) > 450 msec | 5 | 2
  QTcB > 500 msec | 2 | 0
  QTcF > 500 msec | 0 | 0
  QTcB Change from Baseline > 30 msec | 28 | 17
  QTcF Change from Baseline > 30 msec | 21 | 11
  QTcB Change from Baseline > 60 msec | 2 | 4
  QTcF Change from Baseline > 60 msec | 1 | 0

25. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Vital Sign Abnormalities During Phase 2
Description: Heart Rate: increase, ≥120 beats per minute (bpm) and ≥15 relative to baseline (RBL); decrease, ≤50 bpm and ≥15 RBL. Systolic BP: increase, ≥180 mmHg and ≥20 RBL; decrease, ≤90 mmHg and ≥20 RBL. Diastolic BP: increase, ≥105 mmHg and ≥15 RBL; decrease, ≤50 mmHg and ≥15 RBL. For patients missing a baseline value, an on-treatment value was considered potentially clinically relevant if the value meets the criterion value.
Time Frame: as for outcome 24
Population: Phase 2 Safety Sample
Measure: Number; unit: Participants
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 292 | 390
Participants
  Systolic Blood Pressure (SBP) - Standing Increase | 2 | 4
  SBP - Standing Decrease | 0 | 4
  SBP - Supine Increase | 1 | 6
  SBP - Supine Decrease | 2 | 4
  SBP - Sitting Increase | 0 | 0
  SBP - Sitting Decrease | 1 | 0
  Diastolic Blood Pressure (DBP) - Standing Increase | 4 | 7
  DBP - Standing Decrease | 0 | 3
  DBP - Supine Increase | 2 | 5
  DBP - Supine Decrease | 1 | 3
  DBP - Sitting Increase | 0 | 3
  DBP - Sitting Decrease | 0 | 0
  Heart Rate - Standing Increase | 0 | 2
  Heart Rate - Standing Decrease | 1 | 0
  Heart Rate - Supine Increase | 0 | 1
  Heart Rate - Supine Decrease | 1 | 1
  Heart Rate - Sitting Increase | 0 | 1
  Heart Rate - Sitting Decrease | 0 | 0
  Weight - Increase | 26 | 46
  Weight - Decrease | 15 | 6

26. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Laboratory Abnormalities During Phase 2
Description: ULN=upper limit of normal; HDL=high density lipoprotein; LDL=low density lipoprotein. Values for ULN are provided by the lab in the database and could be different for each individual patient based on characteristics such as age, gender, or other patient attributes.
Time Frame: as for outcome 24
Population: Phase 2 Safety Sample; n=number of participants with evaluation at time point
Measure: Number; unit: Participants
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 292 | 390
Participants
  Alkaline Phosphatase ≥ 3 x ULN (n=272, 360) | 0 | 0
  Alanine Aminotransferase ≥ 3 x ULN (n=273, 359) | 3 | 6
  Aspartate Aminotransferase ≥ 3 x ULN (n=273, 359) | 0 | 3
  Blood Urea Nitrogen ≥ 30 mg/dL (n=225, 312) | 0 | 7
  Creatine Kinase >= 3 x ULN (n=273, 360) | 6 | 20
  Creatinine ≥ 2.0 mg/dL (n=271, 359) | 1 | 1
  Lactate Dehydrogenase >= 3 x ULN (n=270, 358) | 0 | 0
  Prolactin > ULN (n=231, 306) | 10 | 9
  Bilirubin Total ≥ 2.0 mg/dL (n=n=272, 360) | 2 | 1
  Uric Acid ≥10.5mg/dL(M)/≥8.5mg/dL(F) (n=273, 360) | 10 | 7
  Total Calcium ≤8.2 mg/dL or ≥12 mg/dL (n=273, 360) | 2 | 13
  Chloride Serum ≤90 mEq/L or ≥118 mEq/L(n=273, 360) | 1 | 4
  Potassium Serum ≤2.5 mEq/L/≥6.5 mEq/L(n=271, 358) | 0 | 1
  Sodium Serum ≤126 mEq/L/≥156 mEq/L (n=273, 360) | 0 | 2
  Hematocrit ≤37(M)/≤32(F)+3 pts↓from BL(n=272, 358) | 5 | 4
  Hemoglobin ≤11.5 g/dL(M)/≤9.5 g/dL(F) (n=272, 359) | 8 | 3
  Leukocytes <=2800 mm^3 or >=16000 mm^3(n=272, 358) | 9 | 2
  Eosinophils Relative (Calculated) ≥10%(n=272, 358) | 9 | 12
  Neutrophils Relative (Calculated) ≤15%(n=272, 358) | 0 | 1
  Platelets ≤75,000 mm^3/≥700,000 mm^3 (n=268, 357) | 1 | 0
  Urine Glucose-any glucose in the urine(n=269,357) | 7 | 13
  Urine Protein Increase of ≥ 2 units (n=269, 357) | 10 | 6
  Glucose (Non-fasting) ≥200 mg/dL (n=78, 89) | 2 | 3
  Glucose (Fasting) ≥ 126 mg/dL (n=251, 332) | 42 | 28
  HDL Cholesterol (combined) <40 mg/dL (n=273, 360) | 94 | 131
  HDL Cholesterol (Fasting) <40 mg/dL (n=252, 332) | 85 | 117
  HDL Cholesterol (Non-fasting) <40 mg/dL (n=79, 91) | 20 | 31
  Total Cholesterol (Combined) ≥240 mg/dL(n=273,360) | 37 | 53
  Total Cholesterol (Fasting) ≥240 mg/dL (n=252,332) | 32 | 49
  Total Cholesterol (Non-fasting) ≥240mg/dL(n=79,92) | 7 | 11
  LDL Cholesterol (Combined) ≥160 mg/dL (n=273, 360) | 30 | 47
  LDL Cholesterol (Fasting) ≥160 mg/dL (n=252, 332) | 28 | 44
  LDL Cholesterol (Non-fasting) ≥160 mg/dL (n=79,91) | 4 | 8
  Triglycerides (Combined) ≥ 200 mg/dL (n=273, 360) | 88 | 108
  Triglycerides (Non-Fasting) ≥ 200 mg/dL (n=79, 93) | 25 | 33
  Triglycerides (Fasting) ≥ 200 mg/dL (n=252, 332) | 73 | 85

27. Secondary Outcome: Median Baseline and Change From Baseline in ECG Measurements During Phase 2
Time Frame: Baseline (end of Ph 1), Phase 2 (a 13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout and Confirmation of Partial Nonresponse Phase)
Population: Phase 2 Safety Sample; n= participants with measurement at time point.
Measure: Median (Full Range); unit: msecs
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 223 | 285
msecs
  QTcBazett (QTcB) at Baseline (n=223, 285) | 415.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 412.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  QTcB Change at Phase 2 Endpoint (n=223, 285) | 4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -8.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  QTcB (0.33) at Baseline (n=223, 284) | 403.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 400.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  QTcB(0.33) Change at Phase 2 Endpoint (n=223, 284) | 4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  PR at Baseline (n=222, 284) | 154.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 150.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  PR Change at Phase 2 Endpoint (n=222, 284) | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  RR at Baseline (n=223, 284) | 845.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 870.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  RR Change at Phase 2 Endpoint (n=223, 284) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  QRS at Baseline (n=223, 284) | 90.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 90.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  QRS Change at Phase 2 Endpoint (n=223, 284) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

28. Secondary Outcome: Median Baseline and Change From Baseline in Heart Rate Vital Sign Measurements During Phase 2
Time Frame: as for outcome 27
Population: Phase 2 Safety Sample; n= participants with measurement at time point.
Measure: Median (Full Range); unit: beats per minute
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 286 | 372
beats per minute
  Supine Heart Rate (HR) at Baseline (n=286, 372) | 76.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 74.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Supine HR Change at Phase 2 Endpoint (n=286, 372) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Sitting Heart Rate (HR) at Baseline (n=51, 67) | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 82.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Sitting HR Change at Phase 2 Endpoint (n=51, 67) | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Standing HR at Baseline (n=260, 333) | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Standing HR Change at Phase 2 Endpoint(n=260, 333) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

29. Secondary Outcome: Median Baseline and Change From Baseline in Blood Pressure (BP) Vital Sign Measurements During Phase 2
Time Frame: as for outcome 27
Population: Phase 2 Safety Sample; n= participants with measurement at time point.
Measure: Median (Full Range); unit: mmHg
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 286 | 372
mmHg
  Supine Systolic BP (SBP) at Baseline (n=286, 372) | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Supine SBP Change at Phase 2 Endpoint (n=286, 372) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Supine Diastolic BP (DBP) at Baseline(n=286, 372) | 76.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 77.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Supine DBP Change at Phase 2 Endpoint (n=286, 372) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Sitting SBP at Baseline (n=51, 67) | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Sitting SBP Change at Phase 2 Endpoint (n=51, 67) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Sitting DBP at Baseline (n=51, 67) | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 80.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Sitting DBP Change at Phase 2 Endpoint (n=51, 67) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Standing SBP at Baseline (n=260, 333) | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Standing SBP Change at Phase 2 Endpoint(n=260,333) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Standing DBP at Baseline (n=260, 333) | 78.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Standing DBP Change at Phase 2 Endpoint(n=260,333) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

30. Secondary Outcome: Median Baseline and Change From Baseline in Weight Vital Sign Measurements At Phase 2 Endpoint
Time Frame: Baseline (end of Ph 1), Phase 2 Endpoint. Phase 2 (a 13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout and Confirmation of Partial Nonresponse Phase)
Population: Phase 2 Safety Sample, participants with measurement at time point.
Measure: Median (Full Range); unit: kg
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 218 | 294
kg
  Weight at Baseline | 76.2 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 76.4 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Weight Change at Phase 2 Endpoint | 0.9 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 1.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

31. Secondary Outcome: Median Baseline and Change From Baseline in Body Mass Index (BMI) Vital Sign Measurements at Phase 2 Endpoint
Time Frame: Baseline (end of Ph 1), Phase 2 Endpoint. Phase 2 (13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout, and Confirmation of Partial Nonresponse Phase)
Population: Phase 2 Safety Sample, participants with measurement at time point.
Measure: Median (Full Range); unit: kg/m^2
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 218 | 294
kg/m^2
  BMI at Baseline | 26.9 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 27.2 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  BMI Change at Phase 2 Endpoint | 0.3 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

32. Secondary Outcome: Median Baseline Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Kinase (CK), and Lactate Dehydrogenase (LD), Phase 2 Safety Sample
Time Frame: Baseline
Population: Phase 2 Safety Sample; n=number of participants with evaluation at time point
Measure: Median (Full Range); unit: U/L
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 266 | 347
U/L
  ALP (n=265, 347) | 72.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 64.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  ALT (n=266, 346) | 20.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 17.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  AST (n=266, 346) | 19.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 20.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  CK (n=266, 347) | 79.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 91.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  LD (n=262, 342) | 168.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 173.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

33. Secondary Outcome: Median Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatine Kinase (CK), and Lactate Dehydrogenase (LD) at the End of Phase 2
Time Frame: as for outcome 31
Population: Phase 2 Safety Sample; n=number of participants with evaluation at time point
Measure: Median (Full Range); unit: U/L
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 266 | 347
U/L
  ALP (n=265, 347) | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  ALT (n=266, 346) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  AST (n=266, 346) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  CK (n=266, 347) | -1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  LD (n=262, 342) | -3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

34. Secondary Outcome: Median Baseline and Change From Baseline in Heart Rate Measurements During Phase 2
Time Frame: as for outcome 27
Population: Phase 2 Safety Sample; n= participants with measurement at time point.
Measure: Median (Full Range); unit: msecs
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 223 | 285
msecs
  Heart Rate at Baseline (n=223, 284) | 71.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 69.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Heart Rate Change at Phase 2 Endpoint (n=223, 284) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

35. Secondary Outcome: Median Baseline Blood Urea Nitrogen (BUN), Total Cholesterol-Fasting (TC), Creatine, Glucose, High Density Lipoprotein Cholesterol-Fasting (HDL-C), Low Density Lipoprotein Cholesterol-Fasting (LDL-C), Bilirubin-Total, Triglycerides, and Uric Acid
Time Frame: Baseline
Population: Phase 2 Safety Sample; n=number of participants with evaluation at time point
Measure: Median (Full Range); unit: U/L
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 266 | 347
U/L
  BUN (n=223, 302) | 11.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 13.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  TC (n=245, 318) | 182.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 174.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Creatine (n=263, 343) | 0.900 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.900 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Glucose (n=242, 312) | 92.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 89.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  HDL-C (n=245, 318) | 47.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 45.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  LDL-C (n=245, 318) | 105.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 101.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Bilirubin (n=265, 347) | 0.40 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.40 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Triglycerides (n=245, 318) | 112.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 114.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Uric Acid (n=266, 347) | 5.55 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 5.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

36. Secondary Outcome: Median Change From Baseline in BUN, TC, Creatine, Glucose, HDL-C, LDL-C, Bilirubin-Total, Triglycerides, and Uric Acid at the End of Phase 2
Time Frame: as for outcome 31
Population: Phase 2 Safety Sample; n=number of participants with evaluation at time point
Measure: Median (Full Range); unit: U/L
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 266 | 347
U/L
  BUN (n=223, 302) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  TC (n=245, 318) | -1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 4.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Creatine (n=263, 343) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Glucose (n=242, 312) | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  HDL-C (n=245, 318) | -1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  LDL-C (n=245, 318) | -4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Bilirubin (n=265, 347) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Triglycerides (n=245, 318) | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Uric Acid (n=266, 347) | -0.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

37. Secondary Outcome: Median Baseline Eosinophils (Relative) and Neutrophils (Relative)
Time Frame: Baseline
Population: Phase 2 Safety Sample; n=number of participants with evaluation at time point
Measure: Median (Full Range); unit: percent of total white blood cell count
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 266 | 347
percent of total white blood cell count
  Eosinophils, relative (n=266, 347) | 2.50 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 2.20 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Neutrophils, relative (n=266, 346) | 67.60 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 58.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

38. Secondary Outcome: Median Change From Baseline in Eosinophils (Relative) and Neutrophils (Relative)
Time Frame: Phase 2 Endpoint. Phase 2 (13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout, and Confirmation of Partial Nonresponse Phase)
Population: Phase 2 Safety Sample; n=number of participants with evaluation at time point
Measure: Median (Full Range); unit: percent of total white blood cell count
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 266 | 347
percent of total white blood cell count
  Eosinophils, relative (n=266, 347) | -0.40 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -0.20 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Neutrophils, relative (n=266, 346) | 0.25 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.60 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

39. Secondary Outcome: Median Baseline Hemoglobin
Time Frame: Baseline
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: g/dL
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 266 | 347
g/dL | 13.75 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 13.80 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

40. Secondary Outcome: Median Change From Baseline in Hemoglobin
Time Frame: as for outcome 38
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: g/dL
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 266 | 347
g/dL | 0.05 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

41. Secondary Outcome: Median Baseline Hematocrit
Time Frame: Baseline
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: percentage of total blood volume
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 265 | 344
percentage of total blood volume | 41.30 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 41.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

42. Secondary Outcome: Median Change From Baseline in Hematocrit
Time Frame: as for outcome 38
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: percentage of total blood volume
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 265 | 344
percentage of total blood volume | 0.30 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.20 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

43. Secondary Outcome: Median Baseline Homeostasis Model Assessment 2 (HOMA2)-Percent Beta
Description: HOMA stands for homeostasis model assessment of insulin resistance and beta-cell function. These are model-based calculations that use fasting insulin and glucose concentrations in order to assess pancreatic beta-cell function and insulin resistance. The HOMA2 model assesses beta-cell function (HOMA2-%β) relative to expected normal function (indexed to 100% for normal function) and is based on predictions from experimental human data on the relationship between insulin and glucose in a fasted state. HOMA2-%Beta is a percentage of 'normal function.'
Time Frame: Baseline
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: percentage of 'normal function'
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 58 | 44
percentage of 'normal function' | 99.95 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 118.70 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

44. Secondary Outcome: Median Baseline Homeostasis Model Assessment 2 HOMA2-Insulin Resistance (IR)
Description: HOMA stands for homeostasis model assessment of insulin resistance and beta-cell function. These are model-based calculations that use fasting insulin and glucose concentrations in order to assess pancreatic beta-cell function and insulin resistance. The HOMA2 model assesses insulin resistance (HOMA2-IR) relative to expected normal function (indexed to 1.0 for normal function) and is based on predictions from experimental human data on the relationship between insulin and glucose in a fasted state. HOMA2-IR is a proportion of 'normal function.'
Time Frame: Baseline
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: proportion of 'normal function'
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 58 | 44
proportion of 'normal function' | 1.14 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 1.42 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

45. Secondary Outcome: Median Change From Baseline in Homeostasis Model Assessment 2(HOMA2)-Percent Beta at Phase 2 Endpoint
Description: as for outcome 43
Time Frame: Baseline (end of Ph 1), Phase 2 Endpoint (endpoint of a 13- to 24-week Stability and Maintenance of Stability Phase, which followed a 2- to 8-week Screening, Washout and Confirmation of Partial Nonresponse Phase)
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: percentage of 'normal function'
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 58 | 44
percentage of 'normal function' | 7.70 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 17.05 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

46. Secondary Outcome: Median Change From Baseline in HOMA2 Model Assesses Insulin Resistance (HOMA2-IR) at Phase 2 Endpoint
Description: as for outcome 44
Time Frame: as for outcome 45
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: proportion of 'normal function'
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 58 | 44
proportion of 'normal function' | 0.09 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.15 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

47. Secondary Outcome: Median Baseline Platelet Count
Time Frame: Baseline
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: x10^9 c/L
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 262 | 345
x10^9 c/L | 297.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 226.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

48. Secondary Outcome: Median Change From Baseline in Platelet Count at Phase 2 Endpoint
Time Frame: as for outcome 31
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: x10^9 c/L
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 262 | 345
x10^9 c/L | -4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

49. Secondary Outcome: Median Baseline Prolactin
Time Frame: Baseline
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: ng/dL
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 6 | 8
ng/dL | 10.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 9.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

50. Secondary Outcome: Median Change From Baseline in Prolactin at Phase 2 Endpoint
Time Frame: as for outcome 31
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: ng/dL
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 6 | 8
ng/dL | -2.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

51. Secondary Outcome: Median Baseline Leukocytes
Time Frame: Baseline
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: x10^3 c/L
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 266 | 347
x10^3 c/L | 8.350 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 6.800 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

52. Secondary Outcome: Median Change From Baseline in Leukocytes at Phase 2 Endpoint
Time Frame: as for outcome 31
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Median (Full Range); unit: x10^3 c/L
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 266 | 347
x10^3 c/L | -0.100 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -0.200 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.

53. Secondary Outcome: Baseline Abnormal Involuntary Movement Scale (AIMS)
Description: The AIMS is an assessment of movement dysfunctions. It is a 12-item instrument assessing abnormal involuntary movements associated with antipsychotic drugs and 'spontaneous' motor disturbance related to the illness itself. Scoring the AIMS consists of rating the severity of movement in 3 main anatomic areas (facial/oral, extremities, and trunk), based on a five-point scale (0=none, 4=severe). The AIMS Total Score has a possible range from 0 to 28. Negative change scores indicate improvement in movement dysfunction.
Time Frame: Baseline
Population: Phase 2 Safety Sample, participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 220 | 295
units on a scale | 0.10 (0.042) | 0.08 (0.028)

54. Secondary Outcome: Unadjusted Mean Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) at Phase 2 Endpoint
Description: as for outcome 53
Time Frame: as for outcome 31
Population: Phase 2 Safety Sample, participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 220 | 295
units on a scale | 0.05 (0.056) | 0.04 (0.043)

55. Secondary Outcome: Baseline in Simpson-Angus Scale (SAS) Total Score
Description: The SAS is a 10-item instrument used to evaluate the presence and severity of parkinsonian symptomatology. It is the most commonly used rating scale for Parkinsonism in clinical trials over the past 25 years. The ten items focus on rigidity rather than bradykinesia, and do not assess subjective rigidity or slowness. Items are rated for severity on a 0-4 scale, with definitions given for each anchor point. The total SAS Score has a possible range from 10 to 50.(lower score=less severe). Negative change scores indicate improvement.
Time Frame: Baseline
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 221 | 295
units on a scale | 10.28 (0.054) | 10.30 (0.048)

56. Secondary Outcome: Unadjusted Mean Change From Baseline in Simpson-Angus Scale (SAS) Total Score at Phase 2 Endpoint
Description: The SAS is a 10-item instrument used to evaluate the presence and severity of parkinsonian symptomatology. It is the most commonly used rating scale for Parkinsonism in clinical trials over the past 25 years. The ten items focus on rigidity rather than bradykinesia, and do not assess subjective rigidity or slowness. Items are rated for severity on a 0-4 scale, with definitions given for each anchor point. The total SAS Score has a possible range from 10 to 50(lower score=less severe). Negative change scores indicate improvement.
Time Frame: as for outcome 31
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 221 | 295
units on a scale | 0.44 (0.118) | 0.15 (0.073)

57. Secondary Outcome: Baseline in Barnes Akathisia Global Clinical Assessment
Description: The Barnes Akathisia Rating Scale is a 4-item scale to assess presence and severity of drug-induced akathisia, including both objective items and subjective items, together with a global clinical assessment of akathisia. Global assessment is made on a scale of 0 to 5 with comprehensive definitions provided for each anchor point on scale: 0=absent; 1=questionable; 2=mild akathisia; 3=moderate akathisia; 4=marked akathisia; 5=severe akathisia. Score has a possible range from 0 (absent) to 5 (severe akathisia). Negative change scores indicate improvement in akathisia.
Time Frame: Baseline
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 221 | 295
units on a scale | 0.09 (0.022) | 0.14 (0.024)

58. Secondary Outcome: Unadjusted Mean Change From Baseline in Barnes Akathisia Global Clinical Assessment at Phase 2 Endpoint
Description: as for outcome 57
Time Frame: as for outcome 31
Population: Phase 2 Safety Sample, number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 221 | 295
units on a scale | 0.14 (0.043) | 0.07 (0.039)

59. Secondary Outcome: Deaths, Treatment-Emergent Serious Adverse Events (SAEs), Adverse Events (AEs) in >=2% of Participants, and AEs Leading to Discontinuation During Phase 3
Description: as for outcome 22
Time Frame: Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: Phase 3 Safety Sample
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 166 | 167
Participants
  Deaths | 1 | 1
  Treatment-Emergent SAEs | 8 | 11
  Treatment-Emergent AEs | 105 | 105
  Treatment-Emergent AEs in >=2% of Participants | 49 | 62
  Treatment-Emergent AEs Leading to Discontinuation | 15 | 19

60. Secondary Outcome: Treatment-Emergent AEs in >=5% of Participants During Phase 3, by Age, Gender, Race, and Maximum Intensity
Description: as for outcome 23
Time Frame: Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: Phase 3 Safety Sample; (n=number of participants in sample for each category)
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 166 | 167
Participants
  Participants <= 50 Years (n=132, 131) | 81 | 84
  Participants >50 Years (n=34, 36) | 24 | 21
  Male Participants (n=70, 81) | 45 | 47
  Female Participants (n=96, 86) | 60 | 58
  White Participants (n=63, 74) | 63 | 74
  Non-White Participants (n=42, 31) | 42 | 31
  Participants with Mild/Grade 1 AE | 75 | 75
  Participants with Moderate/Grade 2 AE | 53 | 55
  Participants with Severe/Grade 3 AE | 11 | 9
  Participants with Very Severe/Grade 4 AE | 1 | 2

61. Secondary Outcome: Participants With Potentially Clinically Relevant Vital Sign Abnormalities During Phase 3
Description: as for outcome 25
Time Frame: Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: Phase 3 Safety Sample; n= number of participants with measurement
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 166 | 167
Participants
  SBP- Standing Increase (n=145, 147) | 0 | 0
  SBP- Standing Decrease (n=145, 147) | 2 | 1
  SBP- Supine Increase (n=165, 164) | 0 | 0
  SBP- Supine Decrease (n=165, 164) | 2 | 2
  SBP- Sitting Increase (n=41, 47) | 0 | 0
  SBP- Sitting Decrease (n=41, 47) | 0 | 1
  DBP- Standing Increase (n=145, 147) | 5 | 1
  DBP- Standing Decrease (n=145, 147) | 0 | 2
  DBP- Supine Increase (n=165, 164) | 4 | 3
  DBP- Supine Decrease (n=165, 164) | 1 | 2
  DBP- Sitting Increase (n=41, 47) | 1 | 0
  DBP- Sitting Decrease (n=41, 47) | 0 | 0
  HR- Standing Increase (n=145, 147) | 1 | 1
  HR- Standing Decrease (n=145, 147) | 2 | 0
  HR- Supine Increase (n=165, 164) | 0 | 0
  HR- Supine Decrease (n=165, 164) | 1 | 1
  HR- Sitting Increase (n=41, 47) | 0 | 0
  HR- Sitting Decrease (n=41, 47) | 0 | 1

62. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Values in Supine Systolic BP During Phase 3
Time Frame: Baseline, During Phase 3 (for highest/lowest values), Week 52
Population: Phase 3 Safety Sample, Week 52 Last Observation Carried Forward (LOCF)
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 162 | 161
mm Hg
  Baseline | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 (LOCF) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Change Value During Phase 3 | 8.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Change Value During Phase 3 | -6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -8.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Baseline Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.640, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.423, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.297, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Lowest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.707, Wilcoxon Rank Sum Test

63. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Values in Supine Diastolic BP During Phase 3
Time Frame: Baseline, During Phase 3 (for highest/lowest values), Week 52
Population: Phase 3 Safety Sample, Week 52 Last Observation Carried Forward (LOCF)
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 162 | 161
mm Hg
  Baseline | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 79.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 (LOCF) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Change Value During Phase 3 | 5.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Change Value During Phase 3 | -6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Baseline Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.656, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.045, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.532, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Lowest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.578, Wilcoxon Rank Sum Test

64. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Values in Supine Heart Rate During Phase 3
Time Frame: Baseline, During Phase 3 (for highest/lowest values), Week 52
Population: Phase 3 Safety Sample, Week 52 Last Observation Carried Forward (LOCF)
Measure: Median (Full Range); unit: beats per minute (bpm)
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 162 | 161
beats per minute (bpm)
  Baseline | 74.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 74.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 (LOCF) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Change Value During Phase 3 | 7.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 8.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Change Value During Phase 3 | -5.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -5.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Baseline Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.619, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.868, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.284, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Lowest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.481, Wilcoxon Rank Sum Test

65. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Values in Sitting Systolic BP During Phase 3
Time Frame: Baseline, During Phase 3 (for highest/lowest values), Week 52
Population: Participants in Phase 3 Safety Sample with measurement; Week 52 LOCF
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 33 | 33
mm Hg
  Baseline | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 (LOCF) | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Change Value During Phase 3 | 8.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Change Value During Phase 3 | -3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Baseline Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.184, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.073, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.020, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Lowest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.206, Wilcoxon Rank Sum Test

66. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Values in Sitting Diastolic BP During Phase 3
Time Frame: Baseline, During Phase 3 (for highest/lowest values), Week 52
Population: Participants in Phase 3 Safety Sample with measurement; Week 52 LOCF
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 33 | 33
mm Hg
  Baseline | 80.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 80.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 (LOCF) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Change Value During Phase 3 | 4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Change Value During Phase 3 | -4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Baseline Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.142, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.110, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.022, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Lowest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.542, Wilcoxon Rank Sum Test

67. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Values in Sitting Heart Rate During Phase 3
Time Frame: Baseline, During Phase 3 (for highest/lowest values), Week 52
Population: Participants in Phase 3 Safety Sample with measurement; Week 52 LOCF
Measure: Median (Full Range); unit: beats per minute ?
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 33 | 33
beats per minute ?
  Baseline | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 76.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 (LOCF) | -4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Change Value During Phase 3 | 3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Change Value During Phase 3 | -4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Baseline Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.916, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.707, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.665, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Lowest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.757, Wilcoxon Rank Sum Test

68. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Values in Standing Systolic BP During Phase 3
Time Frame: Baseline, During Phase 3 (for highest/lowest values), Week 52
Population: Participants in Phase 3 Safety Sample with measurement; Week 52 LOCF
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 143 | 143
mm Hg
  Baseline | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 (LOCF) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Change Value During Phase 3 | 8.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Change Value During Phase 3 | -7.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -8.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Baseline Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.871, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.362, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.295, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Lowest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.519, Wilcoxon Rank Sum Test

69. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Values in Standing Diastolic BP During Phase 3
Time Frame: Baseline, During Phase 3 (for highest/lowest values), Week 52
Population: Participants in Phase 3 Safety Sample with measurement; Week 52 LOCF
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 143 | 143
mm Hg
  Baseline | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 (LOCF) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Change Value During Phase 3 | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Change Value During Phase 3 | -6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Baseline Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.935, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.174, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.527, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Lowest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.753, Wilcoxon Rank Sum Test

70. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Values in Standing Heart Rate During Phase 3
Time Frame: Baseline, During Phase 3 (for highest/lowest values), Week 52
Population: Participants in Phase 3 Safety Sample with measurement; Week 52 LOCF
Measure: Median (Full Range); unit: beats per minute
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 143 | 143
beats per minute
  Baseline | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 78.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 (LOCF) | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Change Value During Phase 3 | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 7.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Change Value During Phase 3 | -7.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Baseline Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.850, Wilcoxon Rank Sum Test
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.709, Wilcoxon Rank Sum Test
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.326, Wilcoxon Rank Sum Test
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Lowest Value Treatment Comparison; Aripiprazole/Placebo; Test type: Superiority or Other; p = 0.201, Wilcoxon Rank Sum Test

71. Secondary Outcome: Baseline and Adjusted Mean Change From Baseline in Weight
Time Frame: Baseline, Weeks 12, 24, 36, 52, During Phase 3 (for highest value)
Population: Observed Cases Data Set, Week 52 LOCF; n= number of participants with value at time point
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 161 | 160
kg
  Baseline (n=161, 160) | 81.33 (1.80) | 80.22 (1.79)
  Change at Week 12 (n=129, 121) | -1.00 (0.67) | 0.28 (0.69)
  Change at Week 24 (n=111, 118) | 0.35 (0.53) | 0.13 (0.51)
  Change at Week 36 (n=89, 98) | 0.64 (0.65) | 0.59 (0.60)
  Change at Week 52 (n=85, 95) | 1.66 (0.78) | 1.61 (0.72)
  Change at Week 52 (LOCF) (n=161, 160) | 0.60 (0.49) | 1.07 (0.49)
  Highest Change Value (n=161, 160) | 2.39 (0.42) | 2.35 (0.42)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Week 52 (LOCF) Treatment Difference; Test type: Superiority or Other; p = 0.491, ANOVA/ANCOVA — ANOVA model, controlling for treatment and mood stabilizer, is used for baseline. ANCOVA model, controlling for treatment, mood stabilizer, and baseline value, is used for mean change from baseline; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.87 to 1.81]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Difference; Test type: Superiority or Other; p = 0.945, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-1.21 to 1.12]

72. Secondary Outcome: Number of Participants Showing Relevant Weight Gain During Phase 3
Description: Relevant weight gain: >=7% increase from baseline
Time Frame: Weeks 12, 24, 36, 52, 52 (LOCF), and throughout Phase 3 (for 'at any time' assessment)
Population: Phase 3 Safety Sample; n=number of participants with measurement at time point
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 163 | 164
Participants
  Weight Gain at Week 12 (n=129, 121) | 3 | 6
  Weight Gain at Week 24 (n=111, 118) | 6 | 11
  Weight Gain at Week 36 (n=89, 98) | 16 | 12
  Weight Gain at Week 52 (n=85, 95) | 16 | 18
  Weight Gain at Week 52 (LOCF) (n=161, 160) | 19 | 22
  Weight Gain at Any Time (n=163, 164) | 23 | 29
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Week 12 Treatment Comparison; Test type: Superiority or Other; p = 0.279, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 24 Treatment Comparison; Test type: Superiority or Other; p = 0.247, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Week 36 Treatment Comparison; Test type: Superiority or Other; p = 0.329, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Week 52 Treatment Comparison; Test type: Superiority or Other; p = 0.928, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Week 52 (LOCF) Treatment Comparison; Test type: Superiority or Other; p = 0.584, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.66 to 2.09]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; "At Any Time" Treatment Comparison; Test type: Superiority or Other; p = 0.369, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer; Risk Ratio (RR) = 1.26, 95% CI 2-sided [0.76 to 2.08]

73. Secondary Outcome: Number of Participants Showing Relevant Weight Loss During Phase 3
Description: Relevant weight loss: >=7% decrease from baseline
Time Frame: Weeks 12, 24, 36, 52, 52 (LOCF), and throughout Phase 3 (for 'at any time' assessment)
Population: Phase 3 Safety Sample; n=number of participants with measurement at time point
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 163 | 164
Participants
  Weight Gain at Week 12 (n=129, 121) | 5 | 6
  Weight Gain at Week 24 (n=111, 118) | 7 | 8
  Weight Gain at Week 36 (n=89, 98) | 7 | 8
  Weight Gain at Week 52 (n=85, 95) | 7 | 5
  Weight Gain at Week 52 (LOCF) (n=161, 160) | 13 | 10
  Weight Gain at Any Time (n=163, 164) | 18 | 18
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Week 12 Treatment Comparison; Test type: Superiority or Other; p = 0.685, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 24 Treatment Comparison; Test type: Superiority or Other; p = 0.792, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Week 36 Treatment Comparison; Test type: Superiority or Other; p = 0.805, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Week 52 Treatment Comparison; Test type: Superiority or Other; p = 0.533, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Week 52 (LOCF) Treatment Comparison; Test type: Superiority or Other; p = 0.545, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.35 to 1.74]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; "At Any Time" Treatment Comparison; Test type: Superiority or Other; p = 0.987, Cochran-Mantel-Haenszel — CMH General Association Test controlling for mood stabilizer; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.54 to 1.86]

74. Secondary Outcome: Median Baseline and Change From Baseline in Body Mass Index (BMI) During Phase 3
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 52, Week 52 (LOCF), During Phase 3 (for lowest/highest values)
Population: Phase 3 Safety Sample; n=number of participants with measurement at time point
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 161 | 160
kg/m^2
  Baseline (n=161, 160) | 27.0 [23.7 to 32.3] | 27.9 [24.1 to 31.5]
  Change at Week 12 (n=129, 121) | 0.0 [-0.6 to 0.4] | 0.2 [-0.1 to 0.8]
  Change at Week 24 (n=111, 118) | 0.1 [-0.4 to 0.6] | 0.2 [-0.4 to 0.9]
  Change at Week 36 (n=89, 98) | 0.1 [-0.5 to 0.9] | 0.4 [-0.4 to 1.2]
  Change at Week 52 (n=85, 95) | 0.5 [-0.1 to 1.4] | 0.7 [-0.2 to 1.6]
  Change at Week 52 (LOCF) (n=161, 160) | 0.2 [-0.6 to 0.9] | 0.5 [-0.3 to 1.2]
  Highest Value During Phase 3 (n=161, 160) | 0.4 [0.0 to 1.2] | 0.7 [0.0 to 1.6]
  Lowest Value During Phase 3 (n=161, 160) | -0.4 [-1.0 to 0.1] | -0.1 [-0.9 to 0.3]
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline; Test type: Superiority or Other; p = 0.646, ANOVA/ANCOVA — ANOVA model, controlling for treatment and mood stabilizer, is used for baseline. ANCOVA model on the rank of the change from baseline, controlling for treatment, mood stabilizer, and the rank of baseline is used for change from baseline
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Week 12 Treatment Comparison; Test type: Superiority or Other; p = 0.006, ANOVA/ANCOVA — [p-value comment as in outcome 74, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Week 24 Treatment Comparison; Test type: Superiority or Other; p = 0.485, ANOVA/ANCOVA — [p-value comment as in outcome 74, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Week 36 Treatment Comparison; Test type: Superiority or Other; p = 0.325, ANOVA/ANCOVA — [p-value comment as in outcome 74, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs Aripiprazole; Week 52 Treatment Comparison; Test type: Superiority or Other; p = 0.374, ANOVA/ANCOVA — [p-value comment as in outcome 74, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs Aripiprazole; Week 52 (LOCF) Treatment Comparison; Test type: Superiority or Other; p = 0.064, ANOVA/ANCOVA — [p-value comment as in outcome 74, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs Aripiprazole; Highest Value Treatment Comparison; Test type: Superiority or Other; p = 0.310, ANOVA/ANCOVA — [p-value comment as in outcome 74, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs Aripiprazole; Lowest Value Treatment Comparison; Test type: Superiority or Other; p = 0.046, ANOVA/ANCOVA — [p-value comment as in outcome 74, analysis 1]

75. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Laboratory Abnormalities During Phase 3
Description: ULN=upper limit of normal; Hb=hemoglobin
Time Frame: Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: Phase 3 Safety Sample; n=number of participants with measurement
Measure: Number; unit: participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 166 | 167
participants
  Alkaline Phosphatase ≥ 3 x ULN (n=166,165) | 2 | 0
  Alanine Aminotransferase ≥ 3 x ULN (n=166,165) | 3 | 3
  Aspartate Aminotransferase ≥ 3 x ULN (n=166,165) | 0 | 0
  Blood Urea Nitrogen ≥ 30 mg/dL (n=139, 138) | 3 | 1
  Creatine Kinase (n=166,165) | 8 | 6
  Creatinine ≥ 2.0 mg/dL (n=166,164) | 0 | 1
  Lactate Dehydrogenase (n=166,164) | 0 | 0
  Prolactin > ULN (n=163, 158) | 14 | 14
  Bilirubin Total ≥ 2.0 mg/dL (n=166, 165) | 2 | 3
  Uric Acid≥10.5 mg/dL(M)/≥ 8.5 mg/dL(F)(n=166, 165) | 4 | 7
  Total Calcium ≤8.2 mg/dL or ≥12 mg/dL (n=166, 165) | 4 | 7
  Chloride Serum ≤90 mEq/L or ≥118 mEq/L(n=166, 165) | 1 | 1
  Potassium Serum ≤2.5 or ≥6.5 mEq/L (n=166, 164) | 0 | 3
  Sodium Serum ≤126 or ≥156 mEq/L (n=166, 165) | 1 | 1
  Hematocrit ≤37(M) or ≤32(F)3 poi (n=166, 164) | 7 | 8
  Hb ≤11.5 g/dl (M) / ≤9.5 g/dL (F) (n=166, 164) | 2 | 4
  Leukocytes (n=166, 164) | 5 | 3
  Eosinophils Relative (Calculated) ≥10 (n=166, 164) | 6 | 11
  Neutrophils Relative (Calculated) ≤15 (n=166, 164) | 0 | 0
  Platelet Count (n=165, 162) | 0 | 0
  Urine Glucose (n=166, 165) | 8 | 8
  Urine Protein (n=166, 165) | 5 | 4
  Glucose (non-fasting) (n=38, 28) | 1 | 0
  Glucose (fasting) (n=159, 158) | 26 | 27
  HDL Cholesterol (combined) (n=166, 165) | 81 | 91
  HDL Cholesterol (fasting) (n=160, 159) | 76 | 88
  HDL Cholesterol (non-fasting) (n=38, 27) | 20 | 11
  Total Cholesterol (combined) (n=166, 165) | 28 | 38
  Total Cholesterol (fasting) (n=160, 159) | 27 | 35
  Total Cholesterol (non-fasting) (n=38, 27) | 3 | 7
  LDL Cholesterol (combined) (n=166, 165) | 24 | 23
  LDL Cholesterol (fasting) (n=160, 159) | 24 | 22
  LDL Cholesterol (non-fasting) (n=38, 27) | 1 | 3
  Triglycerides (combined) (n=166, 165) | 59 | 67
  Triglycerides (non-fasting) (n=38, 28) | 16 | 15
  Triglycerides (fasting) (n=160,159) | 48 | 63

76. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Alkaline Phosphatase (ALP), Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: U/L
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
U/L
  Baseline | 60.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 62.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | 1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | 8.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 7.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline ALP; Test type: Superiority or Other; p = 0.331, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in ALP at Week 52 (LOCF); Test type: Superiority or Other; p = 0.353, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison ALP Highest Change Value During Phase 3; Test type: Superiority or Other; p = 0.298, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

77. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in ALT, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: U/L
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
U/L
  Baseline | 19.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 20.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | -1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 5.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline ALT; Test type: Superiority or Other; p = 0.111, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change in ALT at Week 52 (LOCF); Test type: Superiority or Other; p = 0.948, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison ALT Highest Change Value During Phase 3; Test type: Superiority or Other; p = 0.559, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

78. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in AST, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: U/L
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
U/L
  Baseline | 20.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 22.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | 1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | 5.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline AST; Test type: Superiority or Other; p = 0.077, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change in AST at Week 52 (LOCF); Test type: Superiority or Other; p = 0.255, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison AST Highest Change Value During Phase 3; Test type: Superiority or Other; p = 0.918, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

79. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in BUN, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 138 | 135
mg/dL
  Baseline | 11.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 12.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | 3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline BUN; Test type: Superiority or Other; p = 0.118, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in BUN at Week 52 (LOCF); Test type: Superiority or Other; p = 0.532, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison BUN Highest Value of Change During Phase 3; Test type: Superiority or Other; p = 0.169, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

80. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Total Cholesterol (Fasting), Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 158 | 156
mg/dL
  Baseline | 180.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 181.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | 5.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -0.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | 18.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 20.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Total Cholesterol (fasting); Test type: Superiority or Other; p = 0.878, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in Total Cholesterol (fasting) at Week 52 (LOCF); Test type: Superiority or Other; p = 0.544, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Total Cholesterol (fasting) in Phase 3; Test type: Superiority or Other; p = 0.658, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

81. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Creatine Kinase, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: U/L
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
U/L
  Baseline | 82.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 91.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | 5.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | 33.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 28.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Creatine Kinase; Test type: Superiority or Other; p = 0.043, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from baseline in Creatine Kinase at Week 52 (LOCF); Test type: Superiority or Other; p = 0.019, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Creatine Kinase During Phase 3; Test type: Superiority or Other; p = 0.176, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

82. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Creatinine, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 161
mg/dL
  Baseline | 0.900 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.900 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | 0.000 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.000 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | 0.100 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.100 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Creatinine; Test type: Superiority or Other; p = 0.105, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in Creatinine at Week 52 (LOCF); Test type: Superiority or Other; p = 0.634, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Creatinine During Phase 3; Test type: Superiority or Other; p = 0.958, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

83. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Eosinophils (Relative), Phase 3 Safety Sample
Description: The change values reported are the median of (post baseline percentage (of white blood cell count) minus baseline percentage (of white blood cell count).
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: percent of total white blood cell count
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
percent of total white blood cell count
  Baseline | 2.30 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 2.20 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | 0.00 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -0.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | 0.80 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.90 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Eosinophils (relative); Test type: Superiority or Other; p = 0.507, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in Eosinophils (relative) at Week 52 (LOCF); Test type: Superiority or Other; p = 0.834, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Eosinophils (relative) During Phase 3; Test type: Superiority or Other; p = 0.511, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

84. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Glucose (Fasting), Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 157 | 155
mg/dL
  Baseline | 90.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 90.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 7.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Glucose (fasting); Test type: Superiority or Other; p = 0.741, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in Glucose (fasting) at Week 52 (LOCF); Test type: Superiority or Other; p = 0.962, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Change Value in Glucose (fasting) During Phase 3; Test type: Superiority or Other; p = 0.592, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

85. Secondary Outcome: Median Baseline, Change From Baseline, and Lowest Value of Change in Hemoglobin, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for lowest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: g/dL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
g/dL
  Baseline | 13.80 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 14.00 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | -0.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -0.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Value of Change in Phase 3 | -0.50 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -0.60 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Hemoglobin; Test type: Superiority or Other; p = 0.080, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in Hemoglobin at Week 52 (LOCF); Test type: Superiority or Other; p = 0.868, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Lowest Change Value in Hemoglobin During Phase 3; Test type: Superiority or Other; p = 0.299, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

86. Secondary Outcome: Median Baseline, Change From Baseline, and Lowest Value of Change in Hematocrit, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for lowest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: percentage of total blood volume
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
percentage of total blood volume
  Baseline | 41.40 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 42.15 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | -0.40 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -0.30 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Value of Change in Phase 3 | -1.60 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -1.90 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Hematocrit; Test type: Superiority or Other; p = 0.187, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in Hematocrit During Week 52 (LOCF); Test type: Superiority or Other; p = 0.377, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Lowest Value of Change in Hematocrit During Phase 3; Test type: Superiority or Other; p = 0.494, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

87. Secondary Outcome: Median Baseline, Change From Baseline, and Lowest Value of Change in HDL Cholesterol (Fasting), Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for lowest value
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 158 | 156
mg/dL
  Baseline | 46.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 45.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | -1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Value of Change in Phase 3 | -5.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -5.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline HDL Cholesterol (fasting); Test type: Superiority or Other; p = 0.180, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in HDL Cholesterol (fasting) at Week 52 (LOCF); Test type: Superiority or Other; p = 0.950, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Lowest Value of Change in HDL Cholesterol (fasting) During Phase 3; Test type: Superiority or Other; p = 0.342, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

88. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in HOMA2-Percent Beta, Phase 3 Safety Sample
Description: as for outcome 43
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: percentage of 'normal function'
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 36 | 35
percentage of 'normal function'
  Baseline | 120.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 106.90 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | -6.35 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 8.50 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | -10.85 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 5.30 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline HOMA2-Percent Beta; Test type: Superiority or Other; p = 0.349, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in HOMA2-Percent Beta at Week 52 (LOCF); Test type: Superiority or Other; p = 0.624, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value in HOMA2-Percent Beta During Phase 3; Test type: Superiority or Other; p = 0.329, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

89. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in HOMA2-IR, Phase 3 Safety Sample
Description: as for outcome 44
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: proportion of 'normal function'
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 36 | 35
proportion of 'normal function'
  Baseline | 1.24 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 1.06 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | -0.13 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -0.13 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change During Phase 3 | 0.20 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.37 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline HOMA2-IR; Test type: Superiority or Other; p = 0.550, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline in HOMA2-IR at Week 52 (LOCF); Test type: Superiority or Other; p = 0.554, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in HOMA2-IR, Phase 3 Safety Sample; Test type: Superiority or Other; p = 0.870, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

90. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Lactate Dehydrogenase, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: U/L
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 161
U/L
  Baseline | 161.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 171.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change at Week 52 LOCF | 4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change During Phase 3 | 25.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 19.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Lactate Dehydrogenase; Test type: Superiority or Other; p = 0.004, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Lactate Dehydrogenase; Test type: Superiority or Other; p = 0.034, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Lactate Dehydrogenase During Phase 3; Test type: Superiority or Other; p = 0.091, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

91. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Change Value in LDL Cholesterol (Fasting), Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 158 | 156
mg/dL
  Baseline | 104.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 100.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline in Week 52 LOCF | 3.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change During Phase 3 | 16.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 16.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline LDL Cholesterol (fasting); Test type: Superiority or Other; p = 0.808, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline at Week 52 (LOCF); Test type: Superiority or Other; p = 0.507, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Change Value in LDL Cholesterol (fasting); Test type: Superiority or Other; p = 0.948, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

92. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Neutrophils (Relative), Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: percent of total white blood cell count
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
percent of total white blood cell count
  Baseline | 61.55 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 62.60 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Week 52 LOCF | -1.30 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -0.55 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change During Phase 3 | -6.45 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -6.20 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Neutrophils (relative); Test type: Superiority or Other; p = 0.967, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison in change from Baseline in Neutrophils (relative) at Week 52 (LOCF); Test type: Superiority or Other; p = 0.486, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Neutrophils (relative), Phase 3 Safety Sample; Test type: Superiority or Other; p = 0.323, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

93. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Value of Change in Platelet Count, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest/lowest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: x10^9 c/L
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 163 | 160
x10^9 c/L
  Baseline | 252.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 254.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | -1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -3.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change During Phase 3 | 26.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 17.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Value of Change During Phase 3 | -27.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -22.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline in Platelet Count; Test type: Superiority or Other; p = 0.663, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline at Week 52 (LOCF); Test type: Superiority or Other; p = 0.322, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Platelet Count, Phase 3 Safety Sample; Test type: Superiority or Other; p = 0.358, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Treatment Comparison Lowest Value of Change in Platelet Count, Phase 3 Safety Sample; Test type: Superiority or Other; p = 0.541, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

94. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Prolactin, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 154 | 147
ng/mL
  Baseline | 7.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline in Week 52 LOCF | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change During Phase 3 | 3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Prolactin; Test type: Superiority or Other; p = 0.412, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison, Change from Baseline at Week 52 (LOCF); Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Prolactin, Phase 3 Safety Sample; Test type: Superiority or Other; p = 0.004, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

95. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Total Bilirubin, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 161
mg/dL
  Baseline | 0.40 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.40 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | 0.00 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.00 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Phase 3 | 0.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Total Bilirubin; Test type: Superiority or Other; p = 0.630, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline at Week 52 (LOCF); Test type: Superiority or Other; p = 0.675, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Total Bilirubin, Phase 3 Safety Sample; Test type: Superiority or Other; p = 0.592, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

96. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Triglycerides (Fasting), Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 158 | 156
mg/dL
  Baseline | 130.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 134.5 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | 4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change During Phase 3 | 37.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 42.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Triglycerides (fasting); Test type: Superiority or Other; p = 0.273, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline at Week 52 (LOCF); Test type: Superiority or Other; p = 0.489, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Triglycerides (fasting), Phase 3 Safety Sample; Test type: Superiority or Other; p = 0.415, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

97. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Uric Acid, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
mg/dL
  Baseline | 5.50 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 5.75 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | -0.10 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.00 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Uric Acid | 0.65 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.50 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Uric Acid; Test type: Superiority or Other; p = 0.189, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline at Week 52 (LOCF); Test type: Superiority or Other; p = 0.350, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Uric Acid, Phase 3 Safety Sample; Test type: Superiority or Other; p = 0.799, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

98. Secondary Outcome: Median Baseline, Change From Baseline, and Highest and Lowest Value of Change in Leukocytes, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest/lowest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: x 10^3 c/uL
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
x 10^3 c/uL
  Baseline | 6.900 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 7.650 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | 0.150 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -0.100 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change During Phase 3 | 1.100 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 1.100 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Value of Change During Phase 3 | -0.900 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -1.000 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Leukocytes; Test type: Superiority or Other; p = 0.124, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison Change from Baseline at Week 52 (LOCF); Test type: Superiority or Other; p = 0.295, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Highest Value of Change in Leukocytes, Phase 3; Test type: Superiority or Other; p = 0.735, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Lowest Value of Change in Leukocytes, Phase 3; Test type: Superiority or Other; p = 0.505, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

99. Secondary Outcome: Number of Participants With Potentially Clinically Relevant Electrocardiogram (ECG) Abnormalities During Phase 3
Description: as for outcome 24
Time Frame: Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: Phase 3 Safety Sample
Measure: Number; unit: Participants
Arm/Group | Lithium | Valproate
Number analyzed (Participants) | 166 | 167
Participants
  Tachycardia ≥ 120 bpm and ↑ ≥ 15 bpm | 1 | 0
  Bradycardia ≤ 50 bpm and ↓ 15 bpm | 1 | 1
  Sinus Tachycardia (see description) | 1 | 0
  Sinus Bradycardia (see description) | 1 | 1
  SV Premature Beat - not present → present | 1 | 1
  Ventricular Premature Beat - not present → present | 1 | 0
  SV Tachycardia not present → present | 0 | 0
  Ventricular Tachycardia not present → present | 0 | 0
  Atrial Fibrillation (see description) | 0 | 0
  Atrial Flutter not present → present | 0 | 0
  1st Degree AV Block PR ≥0.20 sec and ↑ ≥0.05 sec | 0 | 0
  2nd Degree AV Block not present → present | 0 | 0
  3rd Degree AV Block not present → present | 0 | 0
  Left Bundle Branch Block not present → present | 12 | 9
  Right Bundle Branch Block not present → present | 6 | 3
  Pre-excitation Syndrome not present → present | 0 | 0
  Other Intraventricular Block (see description) | 1 | 0
  Acute Infarction not present → present | 0 | 0
  Subacute (Recent) Infarction not present → present | 1 | 2
  Old Infarction (see description) | 0 | 0
  Myocardial Ischemia not present → present | 1 | 2
  Symmetrical T-Wave Inversion not present → present | 0 | 1
  QTc Bazett (QTcB) > 450 msec | 12 | 15
  QTc Frederica (QTcF) > 450 msec | 5 | 4
  QTcB > 500 msec | 0 | 1
  QTcF > 500 msec | 0 | 1
  QTcB Change from Baseline > 30 msec | 20 | 25
  QTcF Change from Baseline > 30 msec | 10 | 20
  QTcB Change from Baseline > 60 msec | 3 | 4
  QTcF Change from Baseline > 60 msec | 2 | 3

100. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in QT Interval Corrected for Heart Rate (QTc) Bazett, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: msecs
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 139 | 139
msecs
  Baseline | 415.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 410.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | 3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in QTc Bazett | 6.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 12.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline QTc Bazett; Test type: Superiority or Other; p = 0.213, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison, Change from Baseline in QTc Bazett at Week 52 (LOCF); Test type: Superiority or Other; p = 0.708, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in QTc Bazett, Phase 3; Test type: Superiority or Other; p = 0.107, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

101. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in QTc (0.33), Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: msecs
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 139 | 139
msecs
  Baseline | 404.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 400.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | 1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in QTc (0.33) | 3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 10.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline QTc (0.33); Test type: Superiority or Other; p = 0.205, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison, Change from Baseline in QTc (0.33) at Week 52 (LOCF); Test type: Superiority or Other; p = 0.669, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in QTc (0.33), Phase 3; Test type: Superiority or Other; p = 0.072, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

102. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in PR, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: msecs
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 139 | 139
msecs
  Baseline | 155.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 150.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in PR | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline PR; Test type: Superiority or Other; p = 0.012, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison, Change from Baseline in PR at Week 52 (LOCF); Test type: Superiority or Other; p = 0.027, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in PR, Phase 3; Test type: Superiority or Other; p = 0.128, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

103. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in RR, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: msecs
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 139 | 139
msecs
  Baseline | 857.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 870.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | 3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -4.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in RR | 38.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 20.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Value of Change in RR | -15.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -42.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline RR; Test type: Superiority or Other; p = 0.571, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison, Change from Baseline in RR at Week 52 (LOCF); Test type: Superiority or Other; p = 0.353, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in RR, Phase 3 Safety Sample; Test type: Superiority or Other; p = 0.204, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Treatment Comparison Lowest Value of Change in Prolactin, Phase 3 Safety Sample; Test type: Superiority or Other; p = 0.435, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

104. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in QRS, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: msecs
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 139 | 139
msecs
  Baseline | 89.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 90.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in QRS | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline QRS; Test type: Superiority or Other; p = 0.826, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison, Change from Baseline in QRS at Week 52 (LOCF); Test type: Superiority or Other; p = 0.545, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in QRS, Phase 3; Test type: Superiority or Other; p = 0.372, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

105. Secondary Outcome: Adjusted Mean Change From Baseline in Simpson-Angus Scale (SAS) Total Score During Phase 3
Description: The SAS is a 10-item instrument used to evaluate the presence and severity of parkinsonian symptomatology. It is the most commonly used rating scale for Parkinsonism in clinical trials over the past 25 years. The ten items focus on rigidity rather than bradykinesia, and do not assess subjective rigidity or slowness. Items are rated for severity on a 0-4 scale, with definitions given for each anchor point. The total SAS Score has a possible range from 10 to 50(lower scores=less severe). Negative change scores indicate improvement.
Time Frame: Baseline, Weeks 4,8, 12, 24, 36, 52, throughout Phase 3 (for Highest Value of Change)
Population: Phase 3 Safety Sample, OC Data Set and Week 52 LOCF; n=number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Baseline (n=164, 162) | 10.48 (0.09) | 10.50 (0.09)
  Change at Week 4 (n=160, 161) | -0.02 (0.07) | 0.04 (0.07)
  Change at Week 8 (n=151, 145) | -0.13 (0.06) | -0.03 (0.06)
  Change at Week 12 (n=144, 136) | -0.20 (0.05) | -0.10 (0.05)
  Change at Week 24 (n=113, 120) | -0.24 (0.07) | -0.02 (0.06)
  Change at Week 36 (n=97, 104) | -0.26 (0.09) | 0.01 (0.08)
  Change at Week 52 (n=85, 95) | -0.24 (0.08) | -0.07 (0.07)
  Change at Week 52 LOCF (n=164, 162) | -0.20 (0.06) | -0.10 (0.06)
  Highest Value in Change During Phase 3 (n=164,162) | 0.17 (0.10) | 0.53 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Difference; Test type: Superiority or Other; p = 0.235, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.07 to 0.27]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Highest Value in Change Treatment Difference; Test type: Superiority or Other; p = 0.012, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.36, 95% CI 2-sided [0.08 to 0.64]

106. Secondary Outcome: Median Baseline, Change From Baseline, and Highest Value of Change in Heart Rate, Phase 3 Safety Sample
Time Frame: Baseline, Week 52 (LOCF), Throughout Phase 3 (for highest value)
Population: Phase 3 Safety Sample, participants with measurement
Measure: Median (Full Range); unit: bpm
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 139 | 139
bpm
  Baseline | 70.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 69.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Change from Baseline at Week 52 LOCF | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 0.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Highest Value of Change in Heart Rate | 1.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | 3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
  Lowest Value of Change in Heart Rate | -3.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal. | -2.0 [NA to NA] — Values were not prespecified in statistical analysis plan. The purpose of presentation is to flag potential safety signals for further exploration; only medians are presented to help identify direction (and relevance) of any potential safety signal.
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Treatment Comparison Baseline Heart Rate; Test type: Superiority or Other; p = 0.587, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Treatment Comparison, Change from Baseline in Heart Rate at Week 52 (LOCF); Test type: Superiority or Other; p = 0.386, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 3: Comparison: Placebo vs Aripiprazole; Treatment Comparison Highest Value of Change in Heart Rate, Phase 3; Test type: Superiority or Other; p = 0.405, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer
Statistical Analysis 4: Comparison: Placebo vs Aripiprazole; Treatment Comparison Lowest Value of Change in Heart Rate, Phase 3; Test type: Superiority or Other; p = 0.253, Wilcoxon Rank Sum Test — Wilcoxon Rank Sum Test stratified by mood stabilizer

107. Secondary Outcome: Adjusted Mean Change From Baseline in AIMS Total Score During Phase 3
Description: as for outcome 53
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, 52, throughout Phase 3 (for Highest Value of Change)
Population: Phase 3 Safety Sample, OC Data Set and Week 52 LOCF; n=number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Baseline (n=164, 162) | 0.11 (0.05) | 0.14 (0.05)
  Change at Week 4 (n=160, 162) | -0.01 (0.05) | 0.05 (0.04)
  Change at Week 8 (n=151, 145) | 0.11 (0.08) | 0.11 (0.08)
  Change at Week 12 (n=144, 136) | 0.10 (0.07) | -0.01 (0.07)
  Change at Week 24 (n=113, 120) | 0.13 (0.09) | -0.03 (0.08)
  Change at Week 36 (n=97, 105) | 0.08 (0.08) | -0.07 (0.08)
  Change at Week 52 (n=85, 96) | 0.06 (0.08) | -0.02 (0.08)
  Change at Week 52 LOCF (n=164, 162) | 0.01 (0.06) | 0.06 (0.06)
  Highest Value in Change During Phase 3 (n=164,162) | 0.16 (0.10) | 0.28 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Difference; Test type: Superiority or Other; p = 0.514, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.12 to 0.23]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Highest Value of Change Treatment Difference; Test type: Superiority or Other; p = 0.362, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.14 to 0.38]

108. Secondary Outcome: Adjusted Mean Change From Baseline in AIMS Item 8 During Phase 3
Description: The AIMS is an assessment of movement dysfunctions. It is a 12-item instrument assessing abnormal involuntary movements associated with antipsychotic drugs and 'spontaneous' motor disturbance related to the illness itself. Scoring the AIMS consists of rating the severity of movement in 3 main anatomic areas (facial/oral, extremities, and trunk), based on a five-point scale (0=none, 4=severe). AIMS Item 8 Score range from 0 to 4. A negative score signifies improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, 52, throughout Phase 3 (for Highest Value of Change)
Population: Phase 3 Safety Sample, OC Data Set and Week 52 LOCF; n=number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Baseline (n=164, 162) | 0.04 (0.02) | 0.03 (0.02)
  Change at Week 4 (n=160, 162) | -0.01 (0.01) | 0.03 (0.01)
  Change at Week 8 (n=151, 145) | 0.01 (0.02) | 0.02 (0.02)
  Change at Week 12 (n=144, 136) | 0.02 (0.02) | 0.01 (0.02)
  Change at Week 24 (n=113, 120) | 0.02 (0.02) | 0.00 (0.02)
  Change at Week 36 (n=97, 105) | 0.01 (0.02) | -0.00 (0.02)
  Change at Week 52 (n=85, 96) | -0.00 (0.02) | -0.01 (0.02)
  Change at Week 52 LOCF (n=164, 162) | 0.01 (0.02) | 0.01 (0.02)
  Highest Value in Change During Phase 3 (n=164,162) | 0.03 (0.02) | 0.07 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Difference; Test type: Superiority or Other; p = 0.904, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.04 to 0.04]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Highest Value of Change Treatment Difference; Test type: Superiority or Other; p = 0.222, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.03 to 0.11]

109. Secondary Outcome: Adjusted Mean Change From Baseline in AIMS Item 9 During Phase 3
Description: The AIMS is an assessment of movement dysfunctions. It is a 12-item instrument assessing abnormal involuntary movements associated with antipsychotic drugs and 'spontaneous' motor disturbance related to the illness itself. Scoring the AIMS consists of rating the severity of movement in 3 main anatomic areas (facial/oral, extremities, and trunk), based on a five-point scale (0=none, 4=severe). AIMS Item 9 Score range from 0 to 4. A negative score signifies improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, 52, throughout Phase 3 (for Highest Value of Change)
Population: Phase 3 Safety Sample, OC Data Set and Week 52 LOCF; n=number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Baseline (n=164, 162) | 0.01 (0.01) | 0.01 (0.01)
  Change at Week 4 (n=160, 162) | -0.01 (0.01) | 0.01 (0.01)
  Change at Week 8 (n=151, 145) | 0.03 (0.02) | 0.02 (0.02)
  Change at Week 12 (n=144, 136) | 0.03 (0.02) | 0.01 (0.02)
  Change at Week 24 (n=113, 120) | 0.03 (0.02) | 0.01 (0.02)
  Change at Week 36 (n=97, 105) | 0.03 (0.02) | -0.00 (0.02)
  Change at Week 52 (n=85, 96) | 0.02 (0.02) | -0.00 (0.02)
  Change at Week 52 LOCF (n=164, 162) | 0.01 (0.01) | 0.01 (0.01)
  Highest Value in Change During Phase 3 (n=164,162) | 0.04 (0.02) | 0.05 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Difference; Test type: Superiority or Other; p = 0.808, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.03 to 0.04]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Highest Value of Change Treatment Difference; Test type: Superiority or Other; p = 0.771, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model

110. Secondary Outcome: Adjusted Mean Change From Baseline in AIMS Item 10 During Phase 3
Description: The AIMS is an assessment of movement dysfunctions. It is a 12-item instrument assessing abnormal involuntary movements associated with antipsychotic drugs and 'spontaneous' motor disturbance related to the illness itself. Scoring the AIMS consists of rating the severity of movement in 3 main anatomic areas (facial/oral, extremities, and trunk), based on a five-point scale (0=none, 4=severe). AIMS Item 10 Score range from 0 to 4. A negative score signifies improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, 52, throughout Phase 3 (for Highest Value of Change)
Population: Phase 3 Safety Sample, OC Data Set and Week 52 LOCF; n=number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Baseline (n=164, 162) | 0.02 (0.01) | 0.04 (0.01)
  Change at Week 4 (n=160, 162) | -0.00 (0.01) | 0.03 (0.01)
  Change at Week 8 (n=151, 145) | 0.02 (0.02) | 0.01 (0.02)
  Change at Week 12 (n=144, 136) | 0.02 (0.02) | 0.00 (0.02)
  Change at Week 24 (n=113, 120) | 0.05 (0.03) | -0.01 (0.02)
  Change at Week 36 (n=97, 105) | 0.02 (0.02) | -0.02 (0.02)
  Change at Week 52 (n=85, 96) | 0.01 (0.02) | -0.03 (0.02)
  Change at Week 52 LOCF (n=164, 162) | 0.00 (0.01) | -0.01 (0.01)
  Highest Value in Change During Phase 3 (n=164,162) | 0.04 (0.02) | 0.06 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Difference; Test type: Superiority or Other; p = 0.576, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.05 to 0.03]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Highest Value treatment Difference; Test type: Superiority or Other; p = 0.636, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.05 to 0.08]

111. Secondary Outcome: Adjusted Mean Change From Baseline in Barnes Akathisia Global Clinical Assessment During Phase 3
Description: as for outcome 57
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36, 52, throughout Phase 3 (for Highest Value of Change)
Population: Phase 3 Safety Sample, OC Data Set and Week 52 LOCF; n=number of participants with evaluation at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 164 | 162
units on a scale
  Baseline (n=164, 162) | 0.10 (0.04) | 0.16 (0.04)
  Change at Week 4 (n=160, 162) | -0.01 (0.03) | 0.01 (0.03)
  Change at Week 8 (n=151, 144) | -0.06 (0.02) | -0.04 (0.02)
  Change at Week 12 (n=144, 136) | -0.07 (0.03) | -0.03 (0.03)
  Change at Week 24 (n=113, 120) | -0.06 (0.03) | -0.04 (0.03)
  Change at Week 36 (n=97, 104) | -0.09 (0.03) | -0.05 (0.03)
  Change at Week 52 (n=85, 96) | -0.10 (0.03) | -0.07 (0.03)
  Change at Week 52 LOCF (n=164, 162) | -0.06 (0.02) | -0.05 (0.02)
  Highest Value in Change During Phase 3 (n=164,162) | 0.07 (0.04) | 0.11 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Aripiprazole; Week 52 LOCF Treatment Difference; Test type: Superiority or Other; p = 0.774, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.06 to 0.08]
Statistical Analysis 2: Comparison: Placebo vs Aripiprazole; Highest Value of Change, Treatment Difference; Test type: Superiority or Other; p = 0.444, ANOVA/ANCOVA — [p-value comment as in outcome 71, analysis 1]; Means, differences in means, 95% CI for the differences and p-values are based on the ANOVA/ANCOVA model; Median Difference (Final Values) = 0.04, 95% CI 2-sided [-0.06 to 0.14]

112. Secondary Outcome: Number of Participants Taking Concomitant Medications for Potential Treatment of Extrapyramidal Syndrome (EPS) During Phase 3
Time Frame: Phase 3 (A 52-Week Assessment of Relapse Phase following Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: Phase 3 Safety Sample
Measure: Number; unit: participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 166 | 167
participants
  Any EPS Medications | 36 | 40
  Cardiovascular System-Propanolol | 18 | 21
  Nervous System-Benztropine | 10 | 19
  Nervous System-Biperiden | 4 | 2
  Nervous System-Trihexyphenidyl | 11 | 10

113. Secondary Outcome: Extension Phase: Mean Baseline and Mean Change From Baseline in CGI-BP (Mania)
Description: Clinical Global Impression-Bipolar (CGI-BP) assesses global illness severity and change in patients with bipolar disorder. Patients are rated on Change from Preceding Phase (mania, depression and overall bipolar illness) items (also a 7-point scale [1 to 7], with 1 being normal and 7 being very severely ill). A negative change score signifies improvement.
Time Frame: Baseline, Weeks 8, 16, 24, 32, 40, 48, 56, 64, 72 of LTE Phase. LTE Phase (A 72-week Extension Phase [until study unblinding] following Phase 3 [52 weeks], Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: Number of participants analyzed=extension phase participants, observed cases (OC) data set; n=number of participants evaluated at time point
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 19 | 23
units on a scale
  Mean Baseline (N=19, 23) | 1.26 (0.104) | 1.35 (0.102)
  Mean Change at Week 8 (n=19, 23) | -0.26 (0.104) | -0.30 (0.098)
  Mean Change at Week 16 (n=18, 23) | -0.28 (0.109) | -0.30 (0.098)
  Mean Change at Week 24 (n=17, 20) | -0.29 (0.114) | -0.40 (0.112)
  Mean Change at Week 32 (n=15, 15) | 0.00 (0.309) | -0.33 (0.126)
  Mean Change at Week 40 (n=9, 12) | -0.11 (0.111) | -0.33 (0.142)
  Mean Change at Week 48 (n=9, 9) | -0.11 (0.111) | -0.22 (0.147)
  Mean Change at Week 56 (n=5, 9) | 0.00 (0.000) | -0.22 (0.147)
  Mean Change at Week 64 (n=5, 4) | 0.00 (0.000) | 0.00 (0.000)
  Mean Change at Week 72 (n=1, 2) | 0.00 (0.000) | -0.50 (0.500)

114. Secondary Outcome: Extension Phase: Mean Change From Baseline in CGI-BP (Mania) Severity of Illness at Extension Phase Endpoint
Description: as for outcome 113
Time Frame: Baseline, Extension Phase Endpoint. LTE Phase (A 72-week Extension Phase [until study unblinding] following Phase 3 [52 weeks], Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: extension phase participants, last observation carried forward (LOCF)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 19 | 23
units on a scale | -0.05 (0.247) | -0.35 (0.102)

115. Secondary Outcome: Extension Phase: Mean Change From Baseline in CGI-BP Severity of Illness (Depression) at Extension Phase Endpoint
Description: as for outcome 113
Time Frame: as for outcome 114
Population: extension phase participants, last observation carried forward (LOCF)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 19 | 23
units on a scale | -0.16 (0.138) | 0.00 (0.000)

116. Secondary Outcome: Extension Phase: Mean Baseline and Mean Change From Baseline in CGI-BP Severity of Illness (Depression) Through Extension Phase
Description: as for outcome 113
Time Frame: Baseline, Weeks 8, 16, 24, 32, 40, 48, 56, 64, 72. LTE Phase (A 72-week Extension Phase [until study unblinding] following Phase 3 [52 weeks], Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: as for outcome 113
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 19 | 23
units on a scale
  Mean Baseline (N=19, 23) | 1.21 (0.123) | 1.00 (0.000)
  Mean Change at Week 8 (n=19, 23) | -0.11 (0.130) | 0.00 (0.000)
  Mean Change at Week 16 (n=18, 23) | -0.11 (0.137) | 0.00 (0.000)
  Mean Change at Week 24 (n=17, 20) | -0.12 (0.146) | 0.00 (0.000)
  Mean Change at Week 32 (n=15, 15) | -0.20 (0.175) | 0.00 (0.000)
  Mean Change at Week 40 (n=9, 12) | -0.11 (0.200) | 0.00 (0.000)
  Mean Change at Week 48 (n=9, 9) | -0.11 (0.200) | 0.00 (0.000)
  Mean Change at Week 56 (n=5, 9) | -0.20 (0.200) | 0.00 (0.000)
  Mean Change at Week 64 (n=5, 4) | -0.20 (0.200) | 0.00 (0.000)
  Mean Change at Week 72 (n=1, 2) | 0.00 (0.00) | 0.00 (0.000)

117. Secondary Outcome: Extension Phase: Mean Baseline and Mean Change From Baseline in CGI-BP Severity of Illness (Overall) Through Extension Phase
Description: as for outcome 113
Time Frame: as for outcome 116
Population: as for outcome 113
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 19 | 23
units on a scale
  Mean Baseline (N=19, 23) | 1.37 (0.114) | 1.35 (0.102)
  Mean Change at Week 8 (n=19, 23) | -0.26 (0.129) | -0.30 (0.098)
  Mean Change at Week 16 (n=18, 23) | -0.28 (0.135) | -0.30 (0.098)
  Mean Change at Week 24 (n=17, 20) | -0.29 (0.143) | -0.40 (0.112)
  Mean Change at Week 32 (n=15, 15) | -0.07 (0.330) | -0.33 (0.126)
  Mean Change at Week 40 (n=9, 12) | -0.22 (0.222) | -0.33 (0.142)
  Mean Change at Week 48 (n=9, 9) | -0.22 (0.222) | -0.22 (0.147)
  Mean Change at Week 56 (n=5, 9) | -0.20 (0.200) | -0.22 (0.147)
  Mean Change at Week 64 (n=5, 4) | -0.20 (0.200) | 0.00 (0.000)
  Mean Change at Week 72 (n=1, 2) | 0.00 (0.00) | -0.50 (0.500)

118. Secondary Outcome: Extension Phase: Mean Change From Baseline in CGI-BP Severity of Illness (Overall) at Extension Phase Endpoint
Description: as for outcome 113
Time Frame: as for outcome 114
Population: extension phase participants, last observation carried forward (LOCF)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 19 | 23
units on a scale | -0.11 (0.264) | -0.35 (0.102)

119. Secondary Outcome: Extension Phase: Deaths, Adverse Events (AES), Serious Adverse Events (SAEs), and Discontinuations
Description: as for outcome 22
Time Frame: From first day until 30 days after the last dose of double-blind dosing in the Extension Phase (A 72-week Extension Phase [until study unblinding] following Phase 3 [52 weeks], Phase 2 [13 to 24 weeks] and Phase 1 [2 to 8 weeks])
Population: Extension Phase Safety Sample
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 19 | 23
Participants
  Deaths | 0 | 0
  SAEs | 0 | 0
  AEs | 5 | 8
  Discontinuations due to AEs | 1 | 0
  Treatment-related AEs | 2 | 1

120. Secondary Outcome: Extension Phase: Participants With Potentially Clinically Relevant Metabolic Laboratory Abnormalities During Extension Phase
Description: Metabolic abnormalities considered by the investigator as clinically relevant. (Need normal values for each.)
Time Frame: as for outcome 119
Population: Number of Participants Analyzed=Participants in Extension Phase Safety Sample; n=number of participants with evaluation
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 19 | 23
Participants
  Glucose, non-fasting (n=3,1) | 0 | 0
  Glucose, fasting (n=17, 22) | 2 | 3
  HDL Cholesterol, combined (n=18, 22) | 12 | 11
  HDL Cholesterol, fasting (n=17, 22) | 12 | 11
  HDL Cholesterol, non-fasting (n=2, 1) | 0 | 0
  Total Cholesterol, combined (n=18, 22) | 0 | 1
  Total Cholesterol, fasting (n=17, 22) | 0 | 1
  Total Cholesterol, non-fasting (n=2, 1) | 0 | 0
  LDL Cholesterol, combined (n=18, 22) | 1 | 3
  LDL Cholesterol, fasting (n=17, 22) | 1 | 3
  LDL Cholesterol, non-fasting (n=2, 1) | 0 | 0
  Triglycerides, combined (n=18, 22) | 4 | 0
  Triglycerides, fasting (n=17, 22) | 4 | 0
  Triglycerides, non-fasting (n=2, 1) | 0 | 0

121. Secondary Outcome: Extension Phase: Participants With Potentially Clinically Relevant Vital Sign Abnormalities
Description: Vital sign abnormalities considered by the investigator as clinically relevant.
Time Frame: as for outcome 119
Population: Extension Phase Safety Sample
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 19 | 23
Participants
  Systolic Blood Pressure Increase | 0 | 0
  Systolic Blood Pressure Decrease | 0 | 0
  Diastolic Blood Pressure Increase | 0 | 0
  Diastolic Blood Pressure Decrease | 0 | 0
  Heart Rate Increase | 0 | 0
  Heart Rate Decrease | 0 | 0
  Weight Increase | 1 | 7
  Weight Decrease | 2 | 1

122. Secondary Outcome: Extension Phase: Adverse Events (AEs), by Maximum Intensity
Description: as for outcome 23
Time Frame: as for outcome 119
Population: Participants in Extension Phase Safety Sample with AEs
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 19 | 23
Participants
  Mild / Grade 1 | 4 | 7
  Moderate / Grade 2 | 1 | 2
  Severe / Grade 3 | 0 | 0
  Very Severe / Grade 4 | 0 | 0

123. Secondary Outcome: Extension Phase: Participants With Potentially Clinically Relevant Laboratory Abnormalities
Description: Chemistry, hematology, and urinalysis abnormalities considered by the investigator as clinically relevant. Hematocrit: ≤37%(M)/≤32%(F)+3 percentage pts↓from baseline.
Time Frame: as for outcome 119
Population: Participants in Extension Phase Safety Sample with laboratory evaluation
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 18 | 22
Participants
  Creatine Kinase >= 3 x ULN | 1 | 0
  Hematocrit (see description) | 2 | 0
  Hemoglobin ≤11.5 g/dL(M)/≤9.5 g/dL(F) | 2 | 0
  Eosinophils relative (calculated) ≥10% | 2 | 2
  Urine Glucose (any glucose in the urine) | 0 | 2

124. Secondary Outcome: Extension Phase: Participants With Potentially Clinically Relevant ECG Abnormalities
Description: ECG abnormalities considered by the investigator as clinically relevant.Left Bundle Branch Block: Not present at Baseline--> present post-baseline.
Time Frame: as for outcome 119
Population: Participants in Extension Phase Safety Sample with ECG evaluation
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole
Number analyzed (Participants) | 17 | 21
Participants
  Left Bundle Branch Block (see description) | 4 | 1
  QTcB > 450 msec | 1 | 3
  QTcF > 450 msec | 1 | 1
  QTcB Change from Baseline > 30 msec | 3 | 5
  QTcF Change from Baseline > 30 msec | 4 | 3
  QTcB Change from Baseline > 60 msec | 1 | 0
  QTcF Change from Baseline > 60 msec | 1 | 0

ADVERSE EVENTS:
Groups:
- Single-Blind Aripiprazole: Phase 1 (2 to 8 Week Screening, Washout and Confirmation of Partial Nonresponse Phase): lithium: 0.6-1.0 mmol/L or valproate 50-125 µg/ml. Phase 2 (13 to 24 Week Stability and Maintenance of Stability Phase): 10-mg, 15-mg, or 30-mg doses of aripiprazole and lithium: 0.6-1.0 mmol/L or valproate 50-125 µg/ml.
- Double-Blind Placebo: Phase 3 (52 Week Assessment of Relapse Phase): matching placebo oral tablets and lithium: 0.6-1.0 mmol/L or valproate 50-125 µg/ml.
- Double-Blind Aripiprazole: Phase 3 (52 Week Assessment of Relapse Phase): 10-mg, 15-mg, or 30-mg doses of aripiprazole and lithium: 0.6-1.0 mmol/L or valproate 50-125 µg/ml.
- Extension Phase Placebo: Phase 4 (Extension Phase): matching placebo oral tablets and lithium: 0.6-1.0 mmol/L or valproate 50-125 µg/ml.
- Extension Phase Aripiprazole: Phase 4 (Extension Phase): 10-mg, 15-mg, or 30-mg doses of aripiprazole and lithium: 0.6-1.0 mmol/L or valproate 50-125 µg/ml.
Arm/Group | Single-Blind Aripiprazole | Double-Blind Placebo | Double-Blind Aripiprazole | Extension Phase Placebo | Extension Phase Aripiprazole
Serious Adverse Events (participants affected / at risk) | 15/682 | 8/166 | 11/167 | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 402/682 | 61/166 | 68/167 | 5/19 | 6/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Blind Aripiprazole (N=682) | Double-Blind Placebo (N=166) | Double-Blind Aripiprazole (N=167) | Extension Phase Placebo (N=19) | Extension Phase Aripiprazole (N=23)
MANIA (Psychiatric disorders) | 0 | 2 | 2 | 0 | 0
AGITATION (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
AGGRESSION (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 3 | 2 | 1 | 0 | 0
ALCOHOL ABUSE (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
BIPOLAR DISORDER (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
BIPOLAR I DISORDER (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
HALLUCINATION, VISUAL (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
HALLUCINATION, AUDITORY (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
RADIAL NERVE PALSY (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 2 | 1 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
GASTRITIS VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
BARTHOLIN'S CYST (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 1 | 0 | 0 | 0 | 0
DECAPITATION (General disorders) | 0 | 0 | 1 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 0 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single-Blind Aripiprazole (N=682) | Double-Blind Placebo (N=166) | Double-Blind Aripiprazole (N=167) | Extension Phase Placebo (N=19) | Extension Phase Aripiprazole (N=23)
WEIGHT INCREASED (Investigations) | 28 | 11 | 15 | 0 | 1
INSOMNIA (Psychiatric disorders) | 61 | 16 | 9 | 0 | 2
MOOD ALTERED (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0
RESTLESSNESS (Psychiatric disorders) | 36 | 0 | 2 | 0 | 0
TREMOR (Nervous system disorders) | 94 | 4 | 10 | 0 | 1
HEADACHE (Nervous system disorders) | 61 | 18 | 22 | 1 | 1
SEDATION (Nervous system disorders) | 40 | 0 | 1 | 0 | 0
AKATHISIA (Nervous system disorders) | 99 | 3 | 6 | 0 | 0
DIZZINESS (Nervous system disorders) | 43 | 3 | 7 | 0 | 0
SOMNOLENCE (Nervous system disorders) | 53 | 3 | 1 | 0 | 0
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 37 | 1 | 5 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 60 | 4 | 5 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 39 | 6 | 7 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 0
ANAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 3 | 2 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 1 | 0
PYREXIA (General disorders) | 13 | 5 | 7 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.